

Title: Specified Drug-Use Survey ("Long-Term Use Survey") on Zacras Combination Tablets LD & HD

NCT Number: NCT02181816

Statistical analysis plan Approve Date: 29-Nov-2017

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).

Note; This document was translated into English as the language on original version was Japanese.

# Statistical Analysis Plan Specified Drug-Use Survey ("Long-Term Use Survey") on Zacras Combination Tablets LD & HD



3rd edition prepared on 29 November 2017

# Table of Contents

| 1.0 | Definitions of Terms, etc. and Handling of Test/Measurement Data | |
|---|---|---|
| 1.1 | Definitions | 4 |
| 1.2 | Number of Digits to be Displayed | |
| 1.3 | Level of Significance, Confidence Coefficient | |
| 1.4 | Handling of Test/Measurement Data | |
| 2.0 | Disposition of Patients (Patient Composition Diagram) | 16 |
| 3.0 | Patient Demographics and Baseline Characteristics | 17 |
| 4.0 | Treatment Given | 19 |
| 5.0 | Tabulation/Analysis of Safety | 22 |
| 5.1 | Occurrence of Adverse Events and Adverse Drug Reactions/Infections | 22 |
| 5.1 | 1.1 Occurrence of Adverse Events | 22 |
| 5.1 | 1.2 Occurrence of Adverse Drug Reactions/Infections | 22 |
| 5.2 | Occurrence of Adverse Events and Adverse Drug Reactions/Infections in Patients Exclude | d |
| | from Safety Evaluation | 23 |
| 5.2 | 2.1 Occurrence of Adverse Events | 23 |
| 5.2 | 2.2 Occurrence of Adverse Drug Reactions/Infections | 25 |
| 5.3 | Occurrence of Adverse Events and Adverse Drug Reactions/Infections by Seriousness, Time of | f |
| | Onset, and Outcome | 26 |
| 5.3 | Occurrence of Adverse Events by Seriousness, Time of Onset, and Outcome | 26 |
| 5.3 | Occurrence of Adverse Drug Reactions/Infections by Seriousness, Time of Onset, and | |
| | Outcome | 27 |
| 5.4 | Incidence of Adverse Drug Reaction/Infection by Factors Related to Patient Demographics an | d |
| | Baseline Characteristics and Treatment Given. | 28 |
| 5.5 | Listing of Occurrence of Serious Adverse Events and Serious Adverse Dru | g |
| | Reactions/Infections | 30 |
| 5.5 | 5.1 Occurrence of Serious Adverse Events | 30 |
| 5.5 | 5.2 Occurrence of Serious Adverse Drug Reactions/Infections | 30 |
| 5.6 | Listing of Occurrence of Serious Adverse Events and Serious Adverse Dru | g |
| | Reactions/Infections in Patients Excluded from Safety Evaluation | 31 |
| 5.6 | 6.1 Occurrence of Serious Adverse Events | 31 |
| 5.6 | 6.2 Occurrence of Serious Adverse Drug Reactions/Infections | 32 |
| 5.7 | Changes in Test/Measurement Data over Time | 33 |
| 5.7 | 7.1 Vital Signs (Pulse Rate) | 33 |
| 5.7 | 7.2 Laboratory Tests | 33 |
| 6.0 | Tabulation/Analysis of Efficacy | 34 |
| 6.1 | Changes in Blood Pressure over Time | 34 |
| 6.2 | Changes in Blood Pressure over Time in Patients Who Switch from the Combined Use of | f |
| | Azilsartan and Amlodipine | 34 |

| 6.3 | Changes in Blood Pressure over Time in Patients Except for Those Who Switch from the | |
|---|---|---|
| | Combined Use of Azilsartan and Amlodipine. | 35 |
| 6.4 | Factors that May Affect the Efficacy | 35 |

# 1.0 Definitions of Terms, etc. and Handling of Test/Measurement Data

# 1.1 Definitions

| Term | Definition |
|---|---|
| Zacras | Zacras Combination Tablets are abbreviated as Zacras in this document. |
| SOC | System organ class listed in the MedDRA/J |
| HLGT | High level group term listed in the MedDRA/J |
| PT | Preferred term listed in the MedDRA/J |
| LLT | Lowest level term listed in the MedDRA/J |
| Enrolled patient | Patient allowed to be enrolled |
| Patient from whom the CRF is collected | Patient from whom the CRF has been obtained |
| Patient from whom the CRF is not collected | Enrolled patient from whom the CRF has not been collected |
| Finalized patient | Patient from whom the CRF is collected who has the date of CRF completion entered into the PMS system or who requires no information on the CRF status and has not been excluded from the survey |
| Non-finalized patient | Patient from whom the CRF is collected who has not been finalized |
| Patient included in safety evaluation | Finalized patient who is included in safety evaluation |
| Patient excluded from safety evaluation | Finalized patient who is excluded from safety evaluation |
| Patient included in efficacy evaluation | Patient included in safety evaluation who is included in efficacy evaluation |
| Patient excluded from efficacy evaluation | Patient included in safety evaluation who is excluded from safety evaluation |
| Presence or absence of change in daily dose of Zacras | "Yes" for patients with a change in daily dose between the start of treatment with Zacras and the final assessment |
| Duration of treatment with Zacras | End date of treatment with Zacras - start date of treatment with Zacras + 1 |
| End date of treatment | End date of the final dose described in the column of the end date of |
| | treatment in the CRF; or start date of treatment + 360 days if the end date of |
| | treatment is not described in the CRF and there is a check for "ongoing at 12 |
| | months after the start of treatment with Zacras." |
| Treatment completer | Patient with a duration of treatment with Zacras of ≥ start date of treatment + 360 days |
| Treatment non-completer | Patient with a duration of treatment with Zacras of ≤ start date of treatment + |

| Term | Definition |
|---|---|
| | 359 days |
| Reason for discontinuation | If the duration of treatment with Zacras is $\leq$ start date of treatment + 359 |
| of treatment with Zacras | days, the reason for discontinuation of treatment described in the column of |
| | details on the use of Zacras in the CRF will be employed. |
| | If the duration of treatment with Zacras is $\geq$ start date of treatment + 360 |
| | days, the patient will be handled as a treatment completer; therefore, the |
| | reason for discontinuation of treatment described in the column of details on |
| | the use of Zacras in the CRF will not be employed. |
| Azilsartan and amlodipine | Antihypertensives other than Zacras that are terminated on the start day of |
| besilate (hereinafter referred | treatment with Zacras or the previous day. Antihypertensives other than |
| to as amlodipine) used | Zacras will be classified as described below based on the ingredients and |
| before the start of treatment | their doses listed below. Fixed-dose combinations will also be classified |
| with Zacras | based on individual ingredients and their doses. |
| | Azilsartan 20 mg, amlodipine 2.5 mg, amlodipine 5 mg, combined use of |
| | azilsartan 20 mg/amlodipine 2.5 mg, combined use of azilsartan |
| | 20 mg/amlodipine 5 mg, other |
| Switching to Zacras (by | Switching to Zacras will be classified as described below based on the |
| ingredient/dose) | combination of "azilsartan and amlodipine used before the start of treatment |
| | with Zacras" and "initial dose of Zacras." |
| | Azilsartan 20 mg→Zacras LD, azilsartan 20 mg→Zacras HD, amlodipine |
| | 2.5 mg→Zacras LD, amlodipine 5 mg→Zacras HD, combined use of |
| | azilsartan 20 mg/amlodipine 2.5 mg→Zacras LD, combined use of azilsartan |
| | 20 mg/amlodipine 5 mg→Zacras HD, other |
| Switching to Zacras (by | Switching to Zacras will be classified as described below based on |
| ingredient) | "switching to Zacras (by ingredient/dose)." |
| | "Aazilsartan→Zacras" for "azilsartan 20 mg→Zacras LD" or "azilsartan |
| | 20 mg→Zacras HD" |
| | "Amlodipine→Zacras" for "amlodipine 2.5 mg→Zacras LD" or "amlodipine |
| | 5 mg→Zacras HD" |
| | "Combined use of azilsartan/amlodipine—Zacras" for "combined use of |
| | azilsartan 20 mg/amlodipine 2.5 mg→Zacras LD" or "combined use of |
| | azilsartan 20 mg/amlodipine 5 mg→Zacras HD" "Other" for "other" |
| Dationt who awit-li from | "Other" for "other" Detions with "combined use of exilentar/emledining a Zeeres" for switching |
| Patient who switches from | Patient with "combined use of azilsartan/amlodipine→Zacras" for switching |
| combined use | to Zacras (by ingredient) |

| Term | Definition |
|---|---|
| Duration of disease | (Start date of treatment with Zacras - time of diagnosis of hypertension + 1) |
| | ÷ 365.25. For time of diagnosis of hypertension, 1 will be used as the day, |
| | and January 1 will be used if the month is unknown. The duration of disease |
| | will be handled as missing if the year, month, and day are unknown. |
| ADR, etc. | Abbreviation of "adverse drug reaction/infection" |
| | AE other than those assessed by the investigator to be not related to Zacras |
| | In this document, "adverse drug reaction/infection" is used in titles, and |
| | "adverse drug reaction, etc." is used in the text and tables. |
| SAE | Adverse event assessed by the investigator to be serious |
| | Events included in the MedDRA code list in Takeda Medically Significant |
| | AE List will be handled as serious even if assessed by the investigator to be |
| | non-serious. |
| Number of patients with an | Number of patients who experienced an AE or an ADR, etc. |
| AE or an ADR, etc. | |
| Number of AE or ADR, etc. | Number of reported AE or ADR, etc. |
| Time of onset | Time of onset will be calculated as date of onset of AE (or ADR, etc.) - start |
| | date of treatment + 1. |
| | If the month and day of AE (or ADR, etc.) are unknown, January 1 will be |
| | used for calculation. If an AE (or ADR, etc.) occurs in the same year as |
| | treatment is started, the month and day of starting treatment will be used for |
| | calculation. |
| | If the day of AE (or ADR, etc.) is unknown, 1 will be used for calculation. If |
| | an AE (or ADR, etc.) occurs in the same year and month as treatment is |
| | started, the start date of treatment will be used for calculation. |
| | If the year, month, and day of AE (or ADR, etc.) is unknown, the start date of |
| | treatment will be used for calculation. |
| Patient with concurrent | Patient with a check for diabetes in the column of concurrent illness in the |
| diabetes | CRF or concurrent illness corresponding to Standardised MedDRA query |
| | (hereinafter referred to as SMQ) code 20000041 (hyperglycaemia/new onset |
| | diabetes mellitus SMQ [scope: narrow]) described |
| Patient with concurrent | Patient with a check for dyslipidemia in the column of concurrent illness in |
| dyslipidemia | the CRF or concurrent illness corresponding to SMQ code 20000026 |
| | (dyslipidaemia SMQ [scope: narrow]) described |
| Patient with concurrent | Patient with a check for hyperuricemia in the column of concurrent illness in |
| hyperuricemia | the CRF or concurrent illness corresponding to MedDRA PT code 10020903 |
| | (hyperuricaemia) described |

| Term | Definition |
|---|---|
| Patient with concurrent | Patient with a check for cardiac failure in the column of concurrent illness in |
| cardiac failure | the CRF or concurrent illness corresponding to SMQ code 20000004 |
| | (cardiac failure SMQ [scope: narrow]) described in the column of other |
| | disease: name of disease |
| Patient with concurrent | Patient with a check for myocardial infarction or angina in the column of |
| coronary artery disease | concurrent illness in the CRF, concurrent illness corresponding to SMQ code |
| | 20000043 (ischaemic heart disease SMQ [scope: narrow]) described in the |
| | column of other disease: name of disease, or PT corresponding to SMQ code |
| | 20000047 (myocardial infarction SMQ [scope: narrow]) described in the |
| | column of medical history |
| Patient with concurrent | Patient with a check for myocardial infarction in the column of concurrent |
| myocardial infarction | illness in the CRF or PT corresponding to SMQ code 20000047 (myocardial |
| (including old myocardial | infarction SMQ [scope: narrow]) described in the column of other disease: |
| infarction) | name of disease or medical history |
| Patient with concurrent | Patient with a check for angina in the column of concurrent illness in the |
| angina | CRF or concurrent illness corresponding to MedDRA PT code 10002383 |
| | (angina pectoris), 10002388 (angina unstable), 10036759 (Prinzmetal |
| | angina), or 10058144 (postinfarction angina) described in the column of |
| | other disease: name of disease |
| Patient with concurrent | Patient with concurrent coronary artery disease who is not a patient with |
| coronary artery disease | concurrent myocardial infarction (including old myocardial infarction) or |
| (other) | angina |
| Patient with concurrent atrial | Patient with a check for atrial fibrillation in the column of concurrent illness |
| fibrillation | in the CRF or concurrent illness corresponding to MedDRA PT code |
| | 10003658 (atrial fibrillation) described in the column of other disease: name |
| | of disease |
| Patient with concurrent renal | Patient with a check for chronic kidney disease (CKD), diabetic nephropathy, |
| impairment | nephrosclerosis, or other in the column of concurrent illness in the CRF or |
| | concurrent illness corresponding to the following (1), (2), or (3) described in |
| | the column of other disease: name of disease: |
| | (1) SMQ code 20000213 (chronic kidney disease SMQ [scope: narrow]) |
| | (2) Takeda MedDRA query (hereinafter referred to as TMQ) (Renal |
| | Disease) |
| | (3) TMQ (Renal Impairment) |
| Patient with concurrent | Patient with a check for chronic kidney disease (CKD), diabetic nephropathy, |
| chronic kidney disease | nephrosclerosis, or other in the column of concurrent illness in the CRF or |

| Term | Definition |
|---|---|
| (CKD) | concurrent illness corresponding to SMQ code 20000213 (chronic kidney |
| | disease SMQ [scope: narrow]) described in the column of other disease: |
| | name of disease |
| Patient with concurrent | Patient with a check for diabetic nephropathy in the column of concurrent |
| diabetic nephropathy | illness in the CRF or concurrent illness corresponding to MedDRA PT code |
| | 10061835 (diabetic nephropathy) described in the column of other disease: |
| | name of disease |
| Patient with concurrent | Patient with a check for nephrosclerosis in the column of concurrent illness |
| nephrosclerosis | in the CRF or concurrent illness corresponding to MedDRA PT code |
| | 10029159 (nephrosclerosis) described in the column of other disease: name |
| | of disease |
| Patient with concurrent | Patient with concurrent chronic kidney disease (CKD) who is not a patient |
| chronic kidney disease | with concurrent diabetic nephropathy or nephrosclerosis |
| (CKD) (other) | |
| Patient with concurrent renal | Patient with concurrent renal impairment who is not a patient with |
| impairment (other) | concurrent chronic kidney disease (CKD), diabetic nephropathy, |
| | nephrosclerosis, or chronic kidney disease (CKD) (other) |
| Patient with concurrent | Patient with a check for hepatic steatosis or alcoholic hepatopathy in the |
| hepatic impairment | column of concurrent illness in the CRF or concurrent illness corresponding |
| | to the following (1), (2), or (3) described in the column of other disease: |
| | name of disease: |
| | (1) SMQ code 20000005 (hepatic disorders SMQ [scope: narrow]) |
| | (2) MedDRA PT code 10019708 (hepatic steatosis) |
| | MedDRA PT code 10001627 (alcoholic liver disease) |
| Patient with concurrent | Patient with a check for hepatic steatosis in the column of concurrent illness |
| hepatic steatosis | in the CRF or concurrent illness corresponding to MedDRA PT code |
| | 10019708 (hepatic steatosis) described in the column of other disease: name |
| | of disease |
| Patient with concurrent | Patient with a check for alcoholic hepatopathy in the column of concurrent |
| alcoholic hepatopathy | illness in the CRF or concurrent illness corresponding to MedDRA PT code |
| | 10001627 (alcoholic liver disease) described in the column of other disease: |
| | name of disease |
| Patient with concurrent | Patient with concurrent hepatic impairment who is not a patient with |
| hepatic impairment (other) | concurrent hepatic steatosis or alcoholic hepatopathy |
| Patient with concurrent | Patient with PT corresponding to SMQ code 20000060 (cerebrovascular |
| cerebrovascular disorder | disorders SMQ [scope: narrow]) described in the column of concurrent |

| Term | Definition |
|---|---|
| | illness: other disease: name of disease or medical history in the CRF |
| Age | If the month and day of starting treatment is smaller than the month and day |
| | of birth, age will be calculated as year of starting treatment - year of birth - 1. |
| | If the month and day of starting treatment is equal to or greater than the |
| | month and day of birth, age will be calculated as year of starting treatment - |
| | year of birth. |
| | If the month and day of birth is unknown, January 1 will be used for |
| | calculation. If the day of birth is unknown, 1 will be used for calculation. |
| Young, middle-aged, or | Patient aged 15 years or older and 74 years or younger |
| young-old patient | |
| Old-old patient | Patient aged 75 years or older |
| BMI | BMI will be calculated as body weight (kg) / [0.0001 × height (cm) × height |
| | (cm)]. BMI will be displayed to one decimal place by rounding. |
| Concomitant drug (at the | Concomitant drug that is started before the start of treatment with Zacras and |
| start of treatment with | is not terminated on the day before the start of treatment with Zacras, or |
| Zacras) | concomitant drug that is started on the start day of treatment with Zacras |
| Concomitant drug (during | Concomitant drug used during a period from the start day of treatment with |
| the survey period) | Zacras to the end day of treatment with Zacras |
| Concomitant drug (at the end | Concomitant drug used on the end day of treatment with Zacras |
| of treatment with Zacras) | |
| Antihypertensive used | Drug described in the column for details on the use of other antihypertensive |
| within 2 months before the | in the CRF that is started before the start day of treatment with Zacras and |
| start of treatment with | used within 2 months (60 days) before the start of treatment with Zacras |
| Zacras | (excluding drugs that are started on the start day of treatment with Zacras) |
| Antidiabetic | Drugs with a NHI drug code starting with 396, 2492, or 249941 |
| Antidyslipidemic | Drugs with a NHI drug code starting with 218 or any of the following 7-digit |
| | numbers: |
| | 2190101, 2190102, 2190103, 2190104 |
| Antihyperuricemic | Drugs with a NHI drug code starting with 394 |
| Antihypertensive | ACE inhibitors, angiotensin receptor blockers (ARBs), diuretics (thiazide |
| | and thiazide analogue diuretics), calcium antagonists (hereinafter referred to |
| | as Ca antagonists), direct renin inhibitors, aldosterone |
| | antagonists/potassium-sparing diuretics, vasodilators, β-blockers, central |
| | sympathetic inhibitors, $\alpha\beta$ -blockers, $\alpha_1$ -blockers, fixed-dose combination: |
| | ARB + diuretic, fixed-dose combination: ARB + Ca antagonist, fixed-dose |

| Term | Definition |
|---|---|
| | combination: Ca antagonist + statin, and fixed-dose combination: ARB + Ca |
| | antagonist + diuretic in a list of antihypertensives in the Guidelines for the |
| | Management of Hypertension 2014 (JSH2014) |
| ACE inhibitor | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with the |
| | following 4-digit number: |
| | 2144 |
| | Generic name: captopril, enalapril maleate, perindopril erbumine, lisinopril |
| | hydrate, alacepril, delapril hydrochloride, benazepril hydrochloride, |
| | cilazapril hydrate, imidapril hydrochloride, temocapril hydrochloride, |
| | quinapril hydrochloride, trandolapril |
| ARB | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2149039, 2149040, 2149041, 2149042, 2149044, 2149046, 2149048, |
| | 2149110, 2149111, 2149112, 2149113, 2149119, 2149116, 2149114, |
| | 2149117, 2149118, 2149115, 2149120, 2149122 |
| | Generic name: losartan potassium, candesartan cilexetil, valsartan, |
| | telmisartan, olmesartan medoxomil, irbesartan, azilsartan, losartan |
| | potassium/hydrochlorothiazide, candesartan cilexetil/hydrochlorothiazide, |
| | valsartan/hydrochlorothiazide, telmisartan/hydrochlorothiazide, |
| | irbesartan/trichlormethiazide, candesartan cilexetil/amlodipine besilate, |
| | valsartan/amlodipine besilate, telmisartan/amlodipine besilate, |
| | irbesartan/amlodipine besilate, olmesartan medoxomil/azelnidipine, |
| | valsartan/cilnidipine, azilsartan/amlodipine besilate, telmisartan/amlodipine |
| | besilate/hydrochlorothiazide |
| Diuretic (thiazide and | Drugs described in the column for details on the use of other |
| thiazide analogue diuretic) | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2132003, 2132004, 2132006, 2149103, 2149012, 2135001, 2149007, |
| | 2149003, 2149110, 2149111, 2149112, 2149113, 2149119, 2149122 |
| | Generic name: trichlormethiazide, hydrochlorothiazide, |
| | benzylhydrochlorothiazide, indapamide, mefruside, tripamide, meticrane, |
| | losartan potassium/hydrochlorothiazide, candesartan |
| | cilexetil/hydrochlorothiazide, valsartan/hydrochlorothiazide, |
| | telmisartan/hydrochlorothiazide, irbesartan/trichlormethiazide, |
| | telmisartan/amlodipine besilate/hydrochlorothiazide |

| Term | Definition |
|---|---|
| HCTZ | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2132004, 2149110, 2149111, 2149112, 2149113, 2149122 |
| | Generic name: hydrochlorothiazide, losartan potassium/hydrochlorothiazide, |
| | candesartan cilexetil/hydrochlorothiazide, valsartan/hydrochlorothiazide, |
| | telmisartan/hydrochlorothiazide, telmisartan/amlodipine |
| | besilate/hydrochlorothiazide |
| Dose of HCTZ | The dose of HCTZ is the maximum dose in patients receiving HCTZ. |
| Ca antagonist | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2171022, 2171014, 2171019, 2171020, 2149019, 2149022, 2149043, |
| | 2149027, 2149034, 2149037, 2149038, 2171021, 2149035, 2149030, |
| | 2171006, 2149116, 2149114, 2149117, 2149118, 2149115, 2190101, |
| | 2190102, 2190103, 2190104, 2149120, 2149122 |
| | Generic name: amlodipine besilate, nifedipine, nisoldipine, nitrendipine, |
| | nicardipine hydrochloride, nilvadipine, azelnidipine, manidipine |
| | hydrochloride, efonidipine hydrochloride ethanol, cilnidipine, aranidipine, |
| | benidipine hydrochloride, felodipine, barnidipine hydrochloride, diltiazem |
| | hydrochloride, candesartan cilexetil/amlodipine besilate, |
| | valsartan/amlodipine besilate, telmisartan/amlodipine besilate, |
| | irbesartan/amlodipine besilate, olmesartan medoxomil/azelnidipine, |
| | amlodipine besilate/atorvastatin calcium hydrate, valsartan/cilnidipine, |
| | telmisartan/amlodipine besilate/hydrochlorothiazide |
| Direct renin inhibitor | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with the |
| | following 7-digit number: |
| | 2149047 |
| | Generic name: aliskiren fumarate |
| Aldosterone | Drugs described in the column for details on the use of other |
| antagonist/potassium-sparing | antihypertensive in the CRF that have a NHI drug code starting with any of |
| diuretic | the following 7-digit numbers: |
| | 2133001, 2149045, 2133002 |
| | Generic name: spironolactone, eplerenone, triamterene |
| Aldosterone antagonist | Drugs described in the column for details on the use of other |

| Term | Definition |
|---|---|
| | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2133001, 2149045, |
| | Generic name: spironolactone, eplerenone |
| Potassium-sparing diuretic | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with the |
| | following 7-digit number: |
| | 2133002 |
| | Generic name: triamterene |
| Diuretic | Diuretics (thiazide and thiazide analogue diuretics) or potassium-sparing |
| | diuretics described in the column for details on the use of other |
| | antihypertensive in the CRF |
| Vasodilator | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with the |
| | following 7-digit number: |
| | 2142004 |
| | Generic name: hydralazine hydrochloride |
| β-blocker | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2123011, 2123016, 2149700, 2149031, 2149010, 2123001, 2149029, |
| | 2123008, 2149014, 2149021, 2149028, 2123015, 2123005, 2149025, |
| | 2123009, 2149011 |
| | Generic name: atenolol, bisoprolol fumarate, bisoprolol, betaxolol |
| | hydrochloride, metoprolol tartrate, acebutolol hydrochloride, celiprolol |
| | hydrochloride, propranolol hydrochloride, nipradilol, tilisolol hydrochloride, |
| | nadolol, carteolol hydrochloride, pindolol |
| Central sympathetic inhibitor | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2149001, 2149017, 2145001 |
| | Generic name: clonidine hydrochloride, guanabenz acetate, methyldopa |
| | hydrate |
| αβ-blocker | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |

| Term | Definition |
|---|---|
| | 2149032, 2149018, 2123014, 2149009, 2149036 |
| | Generic name: carvedilol, amosulalol hydrochloride, arotinolol |
| | hydrochloride, labetalol hydrochloride, bevantolol hydrochloride |
| α <sub>1</sub> -blocker | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2149026, 2149015, 2149023, 2149002, 2149020 |
| | Generic name: doxazosin mesilate, bunazosin hydrochloride, terazosin |
| | hydrochloride hydrate, prazosin hydrochloride, urapidil |
| Fixed-dose combination: | Drugs described in the column for details on the use of other |
| ARB + diuretic | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2149110, 2149111, 2149112, 2149113, 2149119, 2149122 |
| | Generic name: losartan potassium/hydrochlorothiazide, candesartan |
| | cilexetil/hydrochlorothiazide, valsartan/hydrochlorothiazide, |
| | telmisartan/hydrochlorothiazide, irbesartan/trichlormethiazide, |
| | telmisartan/amlodipine besilate/hydrochlorothiazide |
| Fixed-dose combination: | Drugs described in the column for details on the use of other |
| ARB + Ca antagonist | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2149116, 2149114, 2149117, 2149118, 2149115, 2149120, 2149122 |
| | Generic name: candesartan cilexetil/amlodipine besilate, |
| | valsartan/amlodipine besilate, telmisartan/amlodipine besilate, |
| | irbesartan/amlodipine besilate, olmesartan medoxomil/azelnidipine, |
| | valsartan/cilnidipine, telmisartan/amlodipine besilate/hydrochlorothiazide |
| Fixed-dose combination: | Drugs described in the column for details on the use of other |
| ARB + Ca antagonist + | antihypertensive in the CRF that have a NHI drug code starting with the |
| diuretic | following 7-digit number: |
| | 2149122 |
| | Generic name: telmisartan/amlodipine besilate/hydrochlorothiazide |
| Fixed-dose combination: Ca | Drugs described in the column for details on the use of other |
| antagonist + statin | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2190101, 2190102, 2190103, 2190104 |
| | Generic name: amlodipine besilate/atorvastatin calcium hydrate |
| Other (antihypertensive) | Vasodilators, $\beta$ -blockers, central sympathetic inhibitors, $\alpha\beta$ -blockers, and |

| Term | Definition |
|---|---|
| | $\alpha_1$ -blockers described in the column for details on the use of other |
| | antihypertensive in the CRF |
| Number of concomitant | The number of drugs described in the column for details on the use of other |
| drugs (antihypertensive other | antihypertensive in the CRF will be tabulated. The fixed-dose combination |
| than Zacras) | will be tabulated as one drug. For instance, "fixed-dose combination: ARB + |
| | diuretic" used concomitantly will be tabulated as one drug. |
| eGFR (mL/min/1.73 m <sup>2</sup> ) | eGFR will be calculated as 194 $\times$ serum creatinine [mg/dL] <sup>-1.094</sup> $\times$ age |
| | [years] <sup>-0.287</sup> (× 0.739 for females). eGFR will be displayed as an integer by |
| | rounding. |
| Summary statistics | Number of patients, mean, standard deviation, minimum, first quartile, |
| | median, third quartile, maximum |

## 1.2 Number of Digits to be Displayed

| Term | Definition |
|---|---|
| Percentage (%) | Incidence of AE or ADR, etc.: |
| | Displayed to two decimal places by rounding |
| | Other: |
| | Displayed to one decimal place by rounding |
| Summary statistics | Mean, median, first quartile, and third quartile: |
| | Displayed to one lower digit than raw data by rounding |
| | Standard deviation: |
| | Displayed to two lower digits than raw data by rounding |
| | Minimum and maximum: |
| | Displayed to the same number of digits as raw data |
| P-value | P-value will be displayed to three decimal places by rounding down. |
| | P-value rounded down to less than 0.001 will be displayed as p<0.001. |

## 1.3 Level of Significance, Confidence Coefficient

Level of significance: 5% (two-sided test)

Confidence coefficient: 95% (two-sided estimate)

## 1.4 Handling of Test/Measurement Data

Test/measurement data will be handled in accordance with the criteria described below (with 1 month as 30 days). If there are multiple pieces of data at the same specified time point, data on the test day closest to the specified day of assessment will be employed, and the latest data among different pieces of data on different days with the same deviation from the specified day of assessment will be

employed. At the final assessment\*, values measured on the day closest to the start date of treatment with Zacras + 374 days will be employed. Values measured 15 days or more after the end day of treatment with Zacras will not be employed.

The number of days from the start day of treatment with Zacras is 1 day for the start day of treatment with Zacras and -1 day for the previous day.

\* After 12 months of treatment with Zacras (or at discontinuation of treatment with Zacras)

| Time point of test | Permissible range (number of days from the start day of treatment) | Specified day of assessment |
|---|---|---|
| At the start of treatment | -90 to 1 | Start date of treatment |
| After 1 month of treatment | 2 to 45 | Start date of treatment + 30 |
| After 2 months of treatment | 46 to 75 | Start date of treatment + 60 |
| After 3 months of treatment | 76 to 105 | Start date of treatment + 90 |
| After 4 months of treatment | 106 to 135 | Start date of treatment + 120 |
| After 5 months of treatment | 136 to 165 | Start date of treatment + 150 |
| After 6 months of treatment | 166 to 195 | Start date of treatment + 180 |
| After 7 months of treatment | 196 to 225 | Start date of treatment + 210 |
| After 8 months of treatment | 226 to 255 | Start date of treatment + 240 |
| After 9 months of treatment | 256 to 285 | Start date of treatment + 270 |
| After 10 months of treatment | 286 to 315 | Start date of treatment + 300 |
| After 11 months of treatment | 316 to 345 | Start date of treatment + 330 |
| After 12 months of treatment | 346 to 375 | Start date of treatment + 360 |
| At the final assessment | 2 to 375 | Start date of treatment + 374 |

#### 2.0 Disposition of Patients (Patient Composition Diagram)

(1) Patients included in tabulation/analysis

**Enrolled patients** 

#### (2) Data tabulated/analyzed

The number of enrolled patients, number of medical institutions involved in patient registration, number of patients from whom the CRF is collected, number of patients from whom the CRF is not collected, number of finalized patients, number of non-finalized patients, number of patients included in safety evaluation, number of patients excluded from safety evaluation, number of patients included in efficacy evaluation, and number of patients excluded from efficacy evaluation will be tabulated.

For the number of medical institutions involved in patient registration, one medical institution with different departments should not be counted more than once.

For patients from whom the CRF is not collected, the number of patients by reason for failure to collect will be tabulated.

For patients excluded from safety evaluation and those excluded from efficacy evaluation, the number of patients by reason for exclusion will be tabulated, and excluded patients will be listed

Patients meeting any of the criteria listed below will be handled as described below regarding whether to employ them or not.

| Criterion | Safety<br>evaluation | Efficacy evaluation |
|---|---|---|
| Prescription before the contract period | × | × |
| [posterior finding] | | |
| Registration 15 days or more after | × | × |
| prescription of Zacras [posterior finding] | | |
| Non-target disease | 0 | × |
| Deviation from exclusion criteria | 0 | × |
| Failure to confirm the intake of Zacras [after | × | × |
| the patient enrollment period] | | |
| Unavailability of follow-up CRF | 0 | 0 |
| It is unknown whether the patient experienced | × | × |
| an AE | | |

o: employed, x: excluded or not employed

#### (3) Table/figure number

Figure 2.0-1, Table 2.0-1

# 3.0 Patient Demographics and Baseline Characteristics

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

# (2) Data tabulated/analyzed

For each variable, patients will be categorized as described below, and the number and proportion of patients will be tabulated.

| Variable | Category |
|---|---|
| Sex | Male, female |
| Age | Summary statistics |
| | <65 years, ≥65 years |
| | <65 years, 65 to <75 years, ≥75 years |
| Duration of disease | <1 year, 1 to <3 years, 3 to <5 years, ≥5 years, unknown |
| Diagnostic category | |
| (at the start of | Outpatient, inpatient |
| treatment with Zacras) | |
| Predisposition to hypersensitivity | No, yes, unknown |
| Concurrent illness | No, yes |
| | Diabetes, dyslipidemia, hyperuricemia, cardiac failure, coronary artery |
| Disposition | disease (myocardial infarction (including old myocardial infarction), |
| (multiple | angina, or other), atrial fibrillation, renal impairment (chronic kidney |
| tabulation) | disease (CKD) [diabetic nephropathy, nephrosclerosis, or other] or |
| uo aiamon) | other), hepatic impairment (hepatic steatosis, alcoholic hepatopathy, or |
| | other), cerebrovascular disorder |
| Medical history | No, yes, unknown |
| Body weight (kg) | Summary statistics |
| | <40, 40 to <50, 50 to <60, 60 to <70, ≥70, not measured |
| BMI (kg/m <sup>2</sup> ) | Summary statistics |
| | <18.5, 18.5 to <25.0, 25.0 to <30.0, ≥30.0, unknown |
| eGFR [at the start of | Summary statistics |
| treatment] | <15, 15 to <30, 30 to <45, 45 to <60, 60 to <90, ≥90, unknown |
| (mL/min/1.73 m <sup>2</sup> ) | 715, 15 to 50, 50 to 715, 15 to 500, 60 to 500, _500, unknown |
| Smoking history | Never smoked, current smoker, past smoker, unknown |
| Drinking history | |
| (drink alcoholic | Yes, no, unknown |
| beverage almost every | |
| day) | |

| Presence or absence | |
|------------------------|---------|
| of breast-feeding (at | |
| the start of treatment | No, yes |
| with Zacras) [only | |
| females] | |

Table 3.0-1

# 4.0 Treatment Given

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

For each variable, patients will be categorized as described below, and the number and

proportion of patients will be tabulated.

| Variable | Category |
|---|---|
| Initial dose of Zacras | LD, HD |
| Presence or absence | |
| of change in daily | No, yes |
| dose of Zacras | |
| | $LD{\rightarrow}HD, HD{\rightarrow}LD, LD{\rightarrow}HD{\rightarrow}LD, HD{\rightarrow}LD{\rightarrow}HD$ |
| Disposition | * This categorization is an example and subject to change depending on |
| | actual data. |
| Duration of treatment | 1 to 180 days, 181 to 360 days, ≥361 days |
| with Zacras | 1 to 100 days, 101 to 300 days, 2301 days |
| Presence or absence | |
| of discontinuation of | No, yes |
| treatment with Zacras | |
| Reason for | Successful achievement of treatment goal, AE, patient's failure to visit |
| discontinuation of | the hospital such as transfer to another hospital, insufficient efficacy, |
| treatment with Zacras | other |
| Azilsartan and | Azilsartan 20 mg, amlodipine 2.5 mg, amlodipine 5 mg, combined use |
| amlodipine used | of azilsartan 20 mg/amlodipine 2.5 mg, combined use of azilsartan |
| before the start of | 20 mg/amlodipine 5 mg, other |
| treatment with Zacras | 20 mg umounpme o mg, outer |
| Switching to Zacras | Azilsartan 20 mg→Zacras LD, azilsartan 20 mg→Zacras HD, |
| (by ingredient/dose) | amlodipine 2.5 mg→Zacras LD, amlodipine 5 mg→Zacras HD, |
| | combined use of azilsartan 20 mg/amlodipine 2.5 mg→Zacras LD, |
| | combined use of azilsartan 20 mg/amlodipine 5 mg→Zacras HD, other |
| Switching to Zacras | Azilsartan→Zacras, amlodipine→Zacras, combined use of |
| (by ingredient) | azilsartan/amlodipine→Zacras, other |
| Treatment with | |
| antihypertensive other | |
| than Zacras (at the | No, yes |
| start of treatment with | |
| Zacras) | |

| <b></b> | |
|---|---|
| Disposition (multiple tabulation)* Antihypertensive other than Zacras: treatment with HCTZ (at the start of treatment with Zacras) | ACE inhibitor, ARB, diuretic (thiazide and thiazide analogue diuretic), Ca antagonist, direct renin inhibitor, aldosterone antagonist, potassium-sparing diuretic, fixed-dose combination: ARB + diuretic, fixed-dose combination: ARB + Ca antagonist, fixed-dose combination: ARB + Ca antagonist + diuretic, fixed-dose combination: Ca antagonist + statin, other |
| Disposition | 6.25 mg, 12.5 mg, other |
| Treatment with antihypertensive other than Zacras (during the survey period) | No, yes |
| Disposition (multiple tabulation)* | ACE inhibitor, ARB, diuretic (thiazide and thiazide analogue diuretic), Ca antagonist, direct renin inhibitor, aldosterone antagonist, potassium-sparing diuretic, fixed-dose combination: ARB + diuretic, fixed-dose combination: ARB + Ca antagonist, fixed-dose combination: ARB + Ca antagonist + diuretic, fixed-dose combination: Ca antagonist + statin, other |
| Antihypertensive other than Zacras: treatment with HCTZ (during the survey period) | No, yes |
| Disposition | 6.25 mg, 12.5 mg, other |
| Treatment with antihypertensive other than Zacras (within 2 months before the start of treatment with Zacras) | No, yes |
| Disposition (multiple tabulation)* | ACE inhibitor, ARB, diuretic (thiazide and thiazide analogue diuretic), Ca antagonist, direct renin inhibitor, aldosterone antagonist, potassium-sparing diuretic, fixed-dose combination: ARB + diuretic, |

| | fixed-dose combination: ARB + Ca antagonist, fixed-dose combination: ARB + Ca antagonist + diuretic, fixed-dose combination: Ca antagonist |
|---|---|
| | + statin, other |
| Number of | |
| concomitant drugs | |
| (antihypertensive | |
| other than Zacras) | |
| (at the start of treatment with Zacras) | $0, 1, 2, 3, 4, 5, \ge 6$ |
| (at the end of treatment with Zacras) | $0, 1, 2, 3, 4, 5, \ge 6$ |
| Concomitant | |
| non-antihypertensive drug (during the survey period) | No, yes |
| Disposition (multiple tabulation) | Antidiabetic, antidyslipidemic, antihyperuricemic, other |

<sup>\*</sup> For fixed-dose combinations, individual ingredients will be tabulated separately. If "fixed-dose combination: ARB + diuretic" is used concomitantly, for instance, "ARB" and "diuretic" will also be tabulated.

Table 4.0-1

# 5.0 Tabulation/Analysis of Safety

## 5.1 Occurrence of Adverse Events and Adverse Drug Reactions/Infections

#### 5.1.1 Occurrence of Adverse Events

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with an AE | Number of patients who experienced an AE |
| Number of AE | Number of reported AE. Multiple episodes of the same AE (PT) in the same patient will be tabulated as the total number of episodes. |
| Incidence of AE | The incidence of AE will be calculated as number of patients with an AE/number of patients included in safety evaluation $\times$ 100. |
| Type of AE | AEs will be classified by SOC and then tabulated by PT. For laboratory tests, AEs will be classified by SOC, then sorted by HLGT, and finally tabulated by PT. For SOC, the number of patients with an AE and the incidence of AE will be listed by SOC internationally agreed order. For PT, the number of patients with an AE and the incidence of AE will be listed in ascending order of PT code. Multiple episodes of the same AE (PT) in the same patient will be tabulated as 1 patient. |

## (3) Table/figure number

Table 5.1-1

## 5.1.2 Occurrence of Adverse Drug Reactions/Infections

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with an ADR, etc. | Number of patients who experienced an ADR, etc. |
| Number of ADR, etc. | Number of reported ADR, etc. Multiple episodes of the same ADR, etc. (PT) in the same patient will be tabulated as the total number of episodes. |
| Incidence of ADR, etc. | The incidence of ADR, etc. will be calculated as number of patients |

| | with an ADR, etc./number of patients included in safety evaluation |
|---|---|
| | × 100. |
| | ADRs, etc. will be classified by SOC and then tabulated by PT. For |
| | laboratory tests, ADRs, etc. will be classified by SOC, then sorted |
| | by HLGT, and finally tabulated by PT. |
| Type of ADR, etc. | For SOC, the number of patients with an ADR, etc. and the |
| | incidence of ADR, etc. will be listed by SOC internationally agreed |
| | order. |
| | For PT, the number of patients with ADR, etc. and the incidence of |
| | ADR, etc. will be listed in ascending order of PT code. Multiple |
| | episodes of the same ADR, etc. (PT) in the same patient will be |
| | tabulated as 1 patient. |

Table 5.1-2

- 5.2 Occurrence of Adverse Events and Adverse Drug Reactions/Infections in Patients Excluded from Safety Evaluation
  - 5.2.1 Occurrence of Adverse Events
    - (1) Patients included in tabulation/analysis

Patients excluded from safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with an AE | Number of patients who experienced an AE |
| Number of AE | Number of reported AE. Multiple episodes of the same AE (PT) in the same patient will be tabulated as the total number of episodes. |
| Incidence of AE | The incidence of AE will be calculated as number of patients with an AE/number of patients excluded from safety evaluation × 100. |
| Type of AE | AEs will be classified by SOC and then tabulated by PT. For laboratory tests, AEs will be classified by SOC, then sorted by HLGT, and finally tabulated by PT. For SOC, the number of patients with an AE and the incidence of AE will be listed by SOC internationally agreed order. For PT, the number of patients with an AE and the incidence of AE will be listed in ascending order of PT code. Multiple episodes of the same AE (PT) in the same patient will be tabulated as 1 patient. |

(3) Table/figure number
Table 5.2-1

# 5.2.2 Occurrence of Adverse Drug Reactions/Infections

(1) Patients included in tabulation/analysis

Patients excluded from safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with an ADR, etc. | Number of patients who experienced an ADR, etc. |
| Number of ADR, etc. | Number of reported ADR, etc. Multiple episodes of the same ADR, etc. (PT) in the same patient will be tabulated as the total number of episodes. |
| Incidence of ADR, etc. | The incidence of ADR, etc. will be calculated as number of patients with an ADR, etc./number of patients excluded from safety evaluation × 100. |
| Type of ADR, etc. | ADRs, etc. will be classified by SOC and then tabulated by PT. For laboratory tests, ADRs, etc. will be classified by SOC, then sorted by HLGT, and finally tabulated by PT. For SOC, the number of patients with an ADR, etc. and the incidence of ADR, etc. will be listed by SOC internationally agreed order. For PT, the number of patients with ADR, etc. and the incidence of ADR, etc. will be listed in ascending order of PT code. Multiple episodes of the same ADR, etc. (PT) in the same patient will be tabulated as 1 patient. |

(3) Table/figure number

Table 5.2-2

- 5.3 Occurrence of Adverse Events and Adverse Drug Reactions/Infections by Seriousness, Time of Onset, and Outcome
  - 5.3.1 Occurrence of Adverse Events by Seriousness, Time of Onset, and Outcome
    - (1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

AEs will be categorized for each variable as described below, and the type of AE will be tabulated.

| Variable | Category |
|---|---|
| Seriousness | Serious, non-serious |
| Time of onset | Days 1 to 180, Days 181 to 360, Day 361 or later |
| Outcome | Recovered, recovering, not recovered, recovered with sequelae, fatal, unknown |

The type of AE will be tabulated as described below.

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients | Number of patients who experienced an AE by SOC/PT |
| Number of AE | Number of reported AE by SOC/PT |
| Type of AE | AEs will be classified by SOC and then tabulated by PT. For |
| | laboratory tests, AEs will be classified by SOC, then sorted by |
| | HLGT, and finally tabulated by PT. |
| | AEs will be listed for SOC by SOC internationally agreed order and |
| | for PT in ascending order of PT code. |
| | Multiple episodes of the same AE (PT) in the same patient will be |
| | tabulated by category as the total number of episodes (for instance, |
| | one episode of serious diarrhoea and one episode of non-serious |
| | diarrhoea in the same patient will be counted once in the respective |
| | categories). |

## (3) Table/figure number

Table 5.3-1

## 5.3.2 Occurrence of Adverse Drug Reactions/Infections by Seriousness, Time of Onset, and Outcome

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

## (2) Data tabulated/analyzed

ADRs, etc. will be categorized for each variable as described below, and the type of ADR will be tabulated.

| Variable | Category |
|---|---|
| Seriousness | Serious, non-serious |
| Time of onset | Days 1 to 180, Days 181 to 360, Day 361 or later |
| Outcome | Recovered, recovering, not recovered, recovered with sequelae, fatal, unknown |

The type of ADR, etc. will be tabulated as described below.

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients | Number of patients who experienced an ADR, etc. by SOC/PT |
| Number of ADR, etc. | Number of reported ADR, etc. by SOC/PT |
| | ADRs, etc. will be classified by SOC and then tabulated by PT. For |
| Type of ADR, etc. | laboratory tests, ADRs, etc. will be classified by SOC, then sorted |
| | by HLGT, and finally tabulated by PT. |
| | ADRs, etc. will be listed for SOC by SOC internationally agreed |
| | order and for PT in ascending order of PT code. |
| | Multiple episodes of the same ADR, etc. (PT) in the same patient |
| | will be tabulated by category as the total number of episodes (for |
| | instance, one episode of serious diarrhoea and one episode of |
| | non-serious diarrhoea in the same patient will be counted once in |
| | the respective categories). |

# (3) Table/figure number

Table 5.3-2

- 5.4 Incidence of Adverse Drug Reaction/Infection by Factors Related to Patient Demographics and Baseline Characteristics and Treatment Given
  - (1) Patients included in tabulation/analysis

    Patients included in safety evaluation

## (2) Data tabulated/analyzed

ADRs, etc. will be categorized for each variable as described below, and the incidence of ADR, etc. will be tabulated.

ADRs, etc. will be categorized for each variable as described below, and the type of ADR, etc. will be tabulated. The type of ADR, etc. will be tabulated as described in Section 5.1. For disposition of treatment with antihypertensive other than Zacras (at the start of treatment with Zacras) and disposition of treatment with antihypertensive other than Zacras (during the survey period), "other" will not be tabulated.

| Variable | Category |
|---|---|
| Sex | Male, female |
| Age | <65 years, ≥65 years |
| | <65 years, 65 to <75 years, ≥75 years |
| Predisposition to | Na |
| hypersensitivity | No, yes, unknown |
| Concurrent illness | No, yes |
| | Diabetes, dyslipidemia, hyperuricemia, cardiac failure, coronary |
| Disposition | artery disease, atrial fibrillation, renal impairment, hepatic |
| | impairment, cerebrovascular disorder |
| Initial dose of Zacras | LD, HD |
| Presence or absence | |
| of change in daily | No, yes |
| dose of Zacras | |
| Switching to Zacras | Azilsartan→Zacras, amlodipine→Zacras, combined use of |
| (by ingredient) | azilsartan/amlodipine→Zacras, other |
| Treatment with | |
| antihypertensive other | |
| than Zacras (at the | No, yes |
| start of treatment with | |
| Zacras) | |
| Disposition (multiple | ACE inhibitor, ARB, diuretic, Ca antagonist, other |
| tabulation)* | ACL minoron, AND, didictic, Ca antagonist, outer |
| Treatment with | No, yes |

| antihypertensive other | |
|------------------------|----------------------------------------------------|
| than Zacras (during | |
| the survey period) | |
| Disposition | ACE inhibitor, ARB, diuretic, Ca antagonist, other |
| (multiple tabulation)* | |

<sup>\*</sup> For fixed-dose combinations, individual ingredients will be tabulated separately. If "fixed-dose combination: ARB + diuretic" is used concomitantly, for instance, "ARB" and "diuretic" will also be tabulated.

Tables 5.4.2-1 to -26

## 5.5 Listing of Occurrence of Serious Adverse Events and Serious Adverse Drug Reactions/Infections

## 5.5.1 Occurrence of Serious Adverse Events

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

## (2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with a SAE | Number of patients who experienced a SAE |
| | Number of reported SAE |
| Number of SAE | Multiple episodes of the same SAE (PT) in the same patient will be |
| | tabulated as the total number of episodes. |
| Incidence of SAE | The incidence of SAE will be calculated as number of patients with |
| Incidence of SAE | a SAE/number of patients included in safety evaluation × 100. |
| | SAEs will be classified by SOC and then tabulated by PT. For |
| | laboratory tests, SAEs will be classified by SOC, then sorted by |
| Type of SAE | HLGT, and finally tabulated by PT. |
| | For SOC, the number of patients with a SAE and the incidence of |
| | SAE will be listed by SOC internationally agreed order. |
| | For PT, the number of patients with a SAE and the incidence of |
| | SAE will be listed in ascending order of PT code. |
| | Multiple episodes of the same SAE (PT) in the same patient will be |
| | tabulated as 1 patient. |
| | The number of patients with a SAE not related to Zacras will be |
| | presented in parentheses. |

## (3) Table/figure number

Table 5.5-1

## 5.5.2 Occurrence of Serious Adverse Drug Reactions/Infections

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with | Number of patients who experienced a serious ADR, etc. |
| a serious ADR, etc. | |
| Number of serious ADR, | Number of reported serious ADR, etc. |

| etc. | Multiple episodes of the same serious ADR, etc. (PT) in the same |
|---|---|
| | patient will be tabulated as the total number of episodes. |
| Incidence of serious ADR, etc. | The incidence of serious ADR, etc. will be calculated as number of patients with a serious ADR, etc./number of patients included in safety evaluation $\times$ 100. |
| Type of serious ADR, etc. | Serious ADRs, etc. will be classified by SOC and then tabulated by PT. For laboratory tests, serious ADRs, etc. will be classified by SOC, then sorted by HLGT, and finally tabulated by PT. For SOC, the number of patients with a serious ADR, etc. and the incidence of serious ADR, etc. will be listed by SOC internationally agreed order. For PT, the number of patients with a serious ADR, etc. and the incidence of serious ADR, etc. will be listed in ascending order of PT code. |

Table 5.5-2

- 5.6 Listing of Occurrence of Serious Adverse Events and Serious Adverse Drug Reactions/Infections in Patients Excluded from Safety Evaluation
  - 5.6.1 Occurrence of Serious Adverse Events
    - (1) Patients included in tabulation/analysis

Patients excluded from safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with a SAE | Number of patients who experienced a SAE |
| Number of SAE | Number of reported SAE |
| | Multiple episodes of the same SAE (PT) in the same patient will |
| | be tabulated as the total number of episodes. |
| Incidence of SAE | The incidence of SAE will be calculated as number of patients |
| | with a SAE/number of patients included in safety evaluation × |
| | 100. |
| Type of SAE | SAEs will be classified by SOC and then tabulated by PT. For |
| | laboratory tests, SAEs will be classified by SOC, then sorted by |
| | HLGT, and finally tabulated by PT. |
| | For SOC, the number of patients with a SAE and the incidence of |

| SAE will be listed by SOC internationally agreed order. |
|-----------------------------------------------------------------|
| For PT, the number of patients with a SAE and the incidence of |
| SAE will be listed in ascending order of PT code. |
| Multiple episodes of the same SAE (PT) in the same patient will |
| be tabulated as 1 patient. |
| The number of patients with a SAE not related to Zacras will be |
| presented in parentheses. |

Table 5.6-1

# 5.6.2 Occurrence of Serious Adverse Drug Reactions/Infections

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with a serious ADR, etc. | Number of patients who experienced a serious ADR, etc. |
| Number of serious ADR, etc. | Number of reported serious ADR, etc. Multiple episodes of the same serious ADR, etc. (PT) in the same patient will be tabulated as the total number of episodes. |
| Incidence of serious ADR, etc. | The incidence of serious ADR, etc. will be calculated as number of patients with a serious ADR, etc./number of patients included in safety evaluation × 100. |
| Type of serious ADR, etc. | Serious ADRs, etc. will be classified by SOC and then tabulated by PT. For laboratory tests, serious ADRs, etc. will be classified by SOC, then sorted by HLGT, and finally tabulated by PT. For SOC, the number of patients with a serious ADR, etc. and the incidence of serious ADR, etc. will be listed by SOC internationally agreed order. For PT, the number of patients with a serious ADR, etc. and the incidence of serious ADR, etc. will be listed in ascending order of PT code. |

# (3) Table/figure number

Table 5.6-2

#### 5.7 Changes in Test/Measurement Data over Time

#### 5.7.1 Vital Signs (Pulse Rate)

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

#### (2) Data tabulated/analyzed

Analyses described below will be performed for patients who have relevant data both before and after treatment with Zacras.

For pulse rate (bpm), summary statistics will be calculated for measured values at each time point of measurement [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment]. For the change from the start of treatment with Zacras, summary statistics will be calculated.

#### (3) Table/figure number

Table 5.7-1

#### 5.7.2 Laboratory Tests

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

#### (2) Data tabulated/analyzed

Analyses described below will be performed for patients who have relevant data both before and after treatment with Zacras.

For white blood cell count, platelet count, AST, ALT,  $\gamma$ -GTP, serum creatinine, BUN, and serum potassium, summary statistics will be calculated for test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment]. For the change from the start of treatment with Zacras, summary statistics will be calculated.

#### (3) Table/figure number

Table 5.7-2

#### 6.0 Tabulation/Analysis of Efficacy

- 6.1 Changes in Blood Pressure over Time
  - (1) Patients included in tabulation/analysis

Patients included in efficacy evaluation

(2) Data tabulated/analyzed

Analyses described below will be performed for patients who have relevant data both before and after treatment with Zacras.

For systolic and diastolic blood pressure, summary statistics and 95% CI for the mean will be calculated for test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment]. The mean and standard deviation of test data will be illustrated.

In addition, the proportion of patients with normal blood pressure at each time point of test will be tabulated. The proportion of patients with normal blood pressure will be illustrated. A patient with normal blood pressure is defined as a patient meeting both criteria listed below. A patient with missing data on systolic and/or diastolic blood pressure will be handled as a patient with missing data.

- •Systolic blood pressure <140 mmHg
- •Diastolic blood pressure <90 mmHg
- (3) Table/figure number

Table 6.1.1, Table 6.1.2, Figure 6.1.1, Figure 6.1.2

- 6.2 Changes in Blood Pressure over Time in Patients Who Switch from the Combined Use of Azilsartan and Amlodipine
  - (1) Patients included in tabulation/analysis

Patients included in efficacy evaluation who switch from combined use

(2) Data tabulated/analyzed

Analyses described below will be performed for patients who have relevant data both before and after treatment with Zacras.

For systolic and diastolic blood pressure, summary statistics and 95% CI for the mean will be calculated for test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment]. For the change from the start of treatment with Zacras, summary statistics and 95% CI for the mean will be calculated. The mean and standard deviation of test data and change will be illustrated. The percentage change from the start of treatment with Zacras ((test data at each time point of test - test data at the start of treatment with Zacras)  $\div$  test data at the start of treatment with Zacras × 100), summary statistics will be calculated. The proportion of patients with normal blood pressure at each time point of test will be tabulated. The proportion of patients with normal blood pressure

will be illustrated.

#### (3) Table/figure number

Table 6.2.1, Table 6.2.2, Table 6.2.3, Figure 6.2.1-1, Figure 6.2.1-2, Figure 6.2.3

- 6.3 Changes in Blood Pressure over Time in Patients Except for Those Who Switch from the Combined Use of Azilsartan and Amlodipine
  - (1) Patients included in tabulation/analysis

Patients included in efficacy evaluation except for those who switch from combined use

(2) Data tabulated/analyzed

Analyses described below will be performed for patients who have relevant data both before and after treatment with Zacras.

For systolic and diastolic blood pressure, summary statistics and 95% CI for the mean will be calculated for test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment]. For the change from the start of treatment with Zacras, summary statistics and 95% CI for the mean will be calculated, and the paired t-test will be performed. The mean and standard deviation of test data and change will be illustrated. For the percentage change from the start of treatment with Zacras, summary statistics will be calculated.

The proportion of patients with normal blood pressure at each time point of test will be tabulated. The proportion of patients with normal blood pressure will be illustrated.

(3) Table/figure number

Table 6.3.1, Table 6.3.2, Table 6.3.3, Figure 6.3.1-1, Figure 6.3.1-2, Figure 6.3.3

- 6.4 Factors that May Affect the Efficacy
  - (1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

Analyses described below will be performed for patients who have relevant data both before and after treatment with Zacras.

For test data on systolic and diastolic blood pressure at the final assessment, summary statistics and 95% CI for the mean will be calculated by the variables listed below.

| Variable | Category |
|--------------------|---------------------------------------|
| Sex | Male, female |
| Age | <65 years, ≥65 years |
| | <65 years, 65 to <75 years, ≥75 years |
| Concurrent illness | No, yes |
| Disposition (multiple tabulation) | Diabetes, dyslipidemia, hyperuricemia, cardiac failure, coronary artery disease, atrial fibrillation, renal impairment, hepatic impairment, cerebrovascular disorder |
|---|---|
| Initial dose of Zacras | LD, HD |
| Presence or absence | |
| of change in daily | No, yes |
| dose of Zacras | |
| Treatment with | |
| antihypertensive other | |
| than Zacras (at the | No, yes |
| start of treatment with | |
| Zacras) | |
| Disposition (multiple tabulation)* | ACE inhibitor, ARB, diuretic, Ca antagonist, other |
| Treatment with | |
| antihypertensive other | No, yes |
| than Zacras (during | 110, 900 |
| the survey period) | |
| Disposition (multiple tabulation)* | ACE inhibitor, ARB, diuretic, Ca antagonist, other |

<sup>\*</sup> For fixed-dose combinations, individual ingredients will be tabulated separately. If "fixed-dose combination: ARB + diuretic" is used concomitantly, for instance, "ARB" and "diuretic" will also be tabulated.

Table 6.4.1

# Statistical Analysis Plan Specified Drug-Use Survey ("Long-Term Use Survey") on Zacras Combination Tablets LD & HD



2nd edition prepared on 16 October 2017

# Table of Contents

| 1.0 | Definitions of Terms, etc. and Handling of Test/Measurement Data | 4 |
|---|---|---|
| 1.1 | Definitions | 4 |
| 1.2 | Number of Digits to be Displayed | |
| 1.3 | Level of Significance, Confidence Coefficient | |
| 1.4 | Handling of Test/Measurement Data | 14 |
| 2.0 | Disposition of Patients (Patient Composition Diagram) | 16 |
| 3.0 | Patient Demographics and Baseline Characteristics | 17 |
| 4.0 | Treatment Given | 19 |
| 5.0 | Tabulation/Analysis of Safety | 22 |
| 5.1 | Occurrence of Adverse Events and Adverse Drug Reactions/Infections | 22 |
| 5.1 | .1 Occurrence of Adverse Events | . 22 |
| 5.1 | .2 Occurrence of Adverse Drug Reactions/Infections | . 22 |
| 5.2 | Occurrence of Adverse Events and Adverse Drug Reactions/Infections in Patients Excluded from | 1 |
| | Safety Evaluation | 23 |
| 5.2 | .1 Occurrence of Adverse Events | 23 |
| 5.2 | .2 Occurrence of Adverse Drug Reactions/Infections | 25 |
| 5.3 | Occurrence of Adverse Events and Adverse Drug Reactions/Infections by Seriousness, Time or | f |
| | Onset, and Outcome | 26 |
| 5.3 | .1 Occurrence of Adverse Events by Seriousness, Time of Onset, and Outcome | 26 |
| 5.3 | .2 Occurrence of Adverse Drug Reactions/Infections by Seriousness, Time of Onset, and Outcome | . 27 |
| 5.4 | Incidence of Adverse Drug Reaction/Infection by Factors Related to Patient Demographics and | l |
| | Baseline Characteristics and Treatment Given | 28 |
| 5.5 | Listing of Occurrence of Serious Adverse Events and Serious Adverse Drug Reactions/Infections | 30 |
| 5.5 | .1 Occurrence of Serious Adverse Events | . 30 |
| 5.5 | .2 Occurrence of Serious Adverse Drug Reactions/Infections | . 30 |
| 5.6 | Listing of Occurrence of Serious Adverse Events and Serious Adverse Drug Reactions/Infections in | 1 |
| | Patients Excluded from Safety Evaluation | 31 |
| 5.6 | .1 Occurrence of Serious Adverse Events | . 31 |
| 5.6 | .2 Occurrence of Serious Adverse Drug Reactions/Infections | . 32 |
| 5.7 | Changes in Test/Measurement Data over Time | 33 |
| 5.7 | .1 Vital Signs (Pulse Rate) | . 33 |
| 5.7 | .2 Laboratory Tests | . 33 |
| 6.0 | Tabulation/Analysis of Efficacy | 34 |
| 6.1 | Changes in Blood Pressure over Time | 34 |
| 6.2 | Changes in Blood Pressure over Time in Patients Who Switch from the Combined Use of Azilsartar | 1 |
| | and Amlodipine | 34 |
| 6.3 | Changes in Blood Pressure over Time in Patients Except for Those Who Switch from the Combined | 1 |
| | Use of Azilsartan and Amlodipine | 35 |

| 6.4 | Factors that May | Affect the Efficacy | <i>y</i> 3 | 5 |
|-----|-------------------|------------------------|------------|---|
| O | i actors that may | Tillett tile Ellitette | , | • |

# 1.0 Definitions of Terms, etc. and Handling of Test/Measurement Data

# 1.1 Definitions

| Term | Definition |
|---|---|
| Zacras | Zacras Combination Tablets are abbreviated as Zacras in this document. |
| SOC | System organ class listed in the MedDRA/J |
| HLGT | High level group term listed in the MedDRA/J |
| PT | Preferred term listed in the MedDRA/J |
| LLT | Lowest level term listed in the MedDRA/J |
| Enrolled patient | Patient allowed to be enrolled |
| Patient from whom the CRF is collected | Patient from whom the CRF has been obtained |
| Patient from whom the CRF is not collected | Enrolled patient from whom the CRF has not been collected |
| Finalized patient | Patient from whom the CRF is collected who has the date of CRF completion entered into the PMS system or who requires no information on the CRF status and has not been excluded from the survey |
| Non-finalized patient | Patient from whom the CRF is collected who has not been finalized |
| Patient included in safety evaluation | Finalized patient who is included in safety evaluation |
| Patient excluded from safety evaluation | Finalized patient who is excluded from safety evaluation |
| Patient included in efficacy evaluation | Patient included in safety evaluation who is included in efficacy evaluation |
| Patient excluded from efficacy evaluation | Patient included in safety evaluation who is excluded from safety evaluation |
| Presence or absence of change in daily dose of Zacras | "Yes" for patients with a change in daily dose between the start of treatment with Zacras and the final assessment |
| Duration of treatment with Zacras | End date of treatment with Zacras - start date of treatment with Zacras + 1 |
| End date of treatment | End date of the final dose described in the column of the end date of |
| | treatment in the CRF; or start date of treatment + 360 days if the end date of |
| | treatment is not described in the CRF and there is a check for "ongoing at 12 |
| | months after the start of treatment with Zacras." |
| Treatment completer | Patient with a duration of treatment with Zacras of ≥ start date of treatment + 360 days |
| Treatment non-completer | Patient with a duration of treatment with Zacras of ≤ start date of treatment + |

| Term | Definition |
|---|---|
| | 359 days |
| Reason for discontinuation | If the duration of treatment with Zacras is $\leq$ start date of treatment + 359 |
| of treatment with Zacras | days, the reason for discontinuation of treatment described in the column of |
| | details on the use of Zacras in the CRF will be employed. |
| | If the duration of treatment with Zacras is $\geq$ start date of treatment + 360 |
| | days, the patient will be handled as a treatment completer; therefore, the |
| | reason for discontinuation of treatment described in the column of details on |
| | the use of Zacras in the CRF will not be employed. |
| Azilsartan and amlodipine | Antihypertensives other than Zacras that are terminated on the start day of |
| besilate (hereinafter referred | treatment with Zacras or the previous day. Antihypertensives other than |
| to as amlodipine) used | Zacras will be classified as described below based on the ingredients and |
| before the start of treatment | their doses listed below. Fixed-dose combinations will also be classified |
| with Zacras | based on individual ingredients and their doses. |
| | Azilsartan 20 mg, amlodipine 2.5 mg, amlodipine 5 mg, combined use of |
| | azilsartan 20 mg/amlodipine 2.5 mg, combined use of azilsartan |
| | 20 mg/amlodipine 5 mg, other |
| Switching to Zacras (by | Switching to Zacras will be classified as described below based on the |
| ingredient/dose) | combination of "azilsartan and amlodipine used before the start of treatment |
| | with Zacras" and "initial dose of Zacras." |
| | Azilsartan 20 mg→Zacras LD, azilsartan 20 mg→Zacras HD, amlodipine |
| | 2.5 mg→Zacras LD, amlodipine 5 mg→Zacras HD, combined use of |
| | azilsartan 20 mg/amlodipine 2.5 mg→Zacras LD, combined use of azilsartan |
| | 20 mg/amlodipine 5 mg→Zacras HD, other |
| Switching to Zacras (by | Switching to Zacras will be classified as described below based on |
| ingredient) | "switching to Zacras (by ingredient/dose)." |
| | "Aazilsartan→Zacras" for "azilsartan 20 mg→Zacras LD" or "azilsartan |
| | 20 mg→Zacras HD" |
| | "Amlodipine→Zacras" for "amlodipine 2.5 mg→Zacras LD" or "amlodipine |
| | 5 mg→Zacras HD" |
| | "Combined use of azilsartan/amlodipine Zacras" for "combined use of |
| | azilsartan 20 mg/amlodipine 2.5 mg→Zacras LD" or "combined use of |
| | azilsartan 20 mg/amlodipine 5 mg→Zacras HD" |
| | "Other" for "other" |
| Patient who switches from | Patient with "combined use of azilsartan/amlodipine→Zacras" for switching |
| combined use | to Zacras (by ingredient) |

| Term | Definition |
|---|---|
| Duration of disease | (Start date of treatment with Zacras - time of diagnosis of hypertension + 1) |
| | $\div$ 365.25. For time of diagnosis of hypertension, 1 will be used as the day, |
| | and January 1 will be used if the month is unknown. The duration of disease |
| | will be handled as missing if the year, month, and day are unknown. |
| ADR, etc. | Abbreviation of "adverse drug reaction/infection" |
| | AE other than those assessed by the investigator to be not related to Zacras |
| | In this document, "adverse drug reaction/infection" is used in titles, and |
| | "adverse drug reaction, etc." is used in the text and tables. |
| SAE | Adverse event assessed by the investigator to be serious |
| | Events included in the MedDRA code list in Takeda Medically Significant |
| | AE List will be handled as serious even if assessed by the investigator to be |
| | non-serious. |
| Number of patients with an | Number of patients who experienced an AE or an ADR, etc. |
| AE or an ADR, etc. | |
| Number of AE or ADR, etc. | Number of reported AE or ADR, etc. |
| Time of onset | Time of onset will be calculated as date of onset of AE (or ADR, etc.) - start |
| | date of treatment + 1. |
| | If the month and day of AE (or ADR, etc.) are unknown, January 1 will be |
| | used for calculation. If an AE (or ADR, etc.) occurs in the same year as |
| | treatment is started, the month and day of starting treatment will be used for |
| | calculation. |
| | If the day of AE (or ADR, etc.) is unknown, 1 will be used for calculation. If |
| | an AE (or ADR, etc.) occurs in the same year and month as treatment is |
| | started, the start date of treatment will be used for calculation. |
| | If the year, month, and day of AE (or ADR, etc.) is unknown, the start date of |
| | treatment will be used for calculation. |
| Patient with concurrent | Patient with a check for diabetes in the column of concurrent illness in the |
| diabetes | CRF or concurrent illness corresponding to Standardised MedDRA query |
| | (hereinafter referred to as SMQ) code 20000041 (hyperglycaemia/new onset |
| | diabetes mellitus SMQ [scope: narrow]) described |
| Patient with concurrent | Patient with a check for dyslipidemia in the column of concurrent illness in |
| dyslipidemia | the CRF or concurrent illness corresponding to SMQ code 20000026 |
| | (dyslipidaemia SMQ [scope: narrow]) described |
| Patient with concurrent | Patient with a check for hyperuricemia in the column of concurrent illness in |
| hyperuricemia | the CRF or concurrent illness corresponding to MedDRA PT code 10020903 |
| | (hyperuricaemia) described |

| Term | Definition |
|---|---|
| Patient with concurrent | Patient with a check for cardiac failure in the column of concurrent illness in |
| cardiac failure | the CRF or concurrent illness corresponding to SMQ code 20000004 |
| | (cardiac failure SMQ [scope: narrow]) described in the column of other |
| | disease: name of disease |
| Patient with concurrent | Patient with a check for myocardial infarction or angina in the column of |
| coronary artery disease | concurrent illness in the CRF, concurrent illness corresponding to SMQ code |
| | 20000043 (ischaemic heart disease SMQ [scope: narrow]) described in the |
| | column of other disease: name of disease, or PT corresponding to SMQ code |
| | 20000047 (myocardial infarction SMQ [scope: narrow]) described in the |
| | column of medical history |
| Patient with concurrent | Patient with a check for myocardial infarction in the column of concurrent |
| myocardial infarction | illness in the CRF or PT corresponding to SMQ code 20000047 (myocardial |
| (including old myocardial | infarction SMQ [scope: narrow]) described in the column of other disease: |
| infarction) | name of disease or medical history |
| Patient with concurrent | Patient with a check for angina in the column of concurrent illness in the |
| angina | CRF or concurrent illness corresponding to MedDRA PT code 10002383 |
| | (angina pectoris), 10002388 (angina unstable), 10036759 (Prinzmetal |
| | angina), or 10058144 (postinfarction angina) described in the column of |
| | other disease: name of disease |
| Patient with concurrent | Patient with concurrent coronary artery disease who is not a patient with |
| coronary artery disease | concurrent myocardial infarction (including old myocardial infarction) or |
| (other) | angina |
| Patient with concurrent atrial | Patient with a check for atrial fibrillation in the column of concurrent illness |
| fibrillation | in the CRF or concurrent illness corresponding to MedDRA PT code |
| | 10003658 (atrial fibrillation) described in the column of other disease: name |
| | of disease |
| Patient with concurrent renal | Patient with a check for chronic kidney disease (CKD), diabetic nephropathy, |
| impairment | nephrosclerosis, or other in the column of concurrent illness in the CRF or |
| | concurrent illness corresponding to the following (1), (2), or (3) described in |
| | the column of other disease: name of disease: |
| | (1) SMQ code 20000213 (chronic kidney disease SMQ [scope: narrow]) |
| | (2) Takeda MedDRA query (hereinafter referred to as TMQ) (Renal |
| | Disease) |
| | (3) TMQ (Renal Impairment) |
| Patient with concurrent | Patient with a check for chronic kidney disease (CKD), diabetic nephropathy, |
| chronic kidney disease | nephrosclerosis, or other in the column of concurrent illness in the CRF or |

| Term | Definition |
|---|---|
| (CKD) | concurrent illness corresponding to SMQ code 20000213 (chronic kidney |
| | disease SMQ [scope: narrow]) described in the column of other disease: |
| | name of disease |
| Patient with concurrent | Patient with a check for diabetic nephropathy in the column of concurrent |
| diabetic nephropathy | illness in the CRF or concurrent illness corresponding to MedDRA PT code |
| | 10061835 (diabetic nephropathy) described in the column of other disease: |
| | name of disease |
| Patient with concurrent | Patient with a check for nephrosclerosis in the column of concurrent illness |
| nephrosclerosis | in the CRF or concurrent illness corresponding to MedDRA PT code |
| | 10029159 (nephrosclerosis) described in the column of other disease: name |
| | of disease |
| Patient with concurrent | Patient with concurrent chronic kidney disease (CKD) who is not a patient |
| chronic kidney disease | with concurrent diabetic nephropathy or nephrosclerosis |
| (CKD) (other) | |
| Patient with concurrent renal | Patient with concurrent renal impairment who is not a patient with |
| impairment (other) | concurrent chronic kidney disease (CKD), diabetic nephropathy, |
| | nephrosclerosis, or chronic kidney disease (CKD) (other) |
| Patient with concurrent | Patient with a check for hepatic steatosis or alcoholic hepatopathy in the |
| hepatic impairment | column of concurrent illness in the CRF or concurrent illness corresponding |
| | to the following (1), (2), or (3) described in the column of other disease: |
| | name of disease: |
| | (1) SMQ code 20000005 (hepatic disorders SMQ [scope: narrow]) |
| | (2) MedDRA PT code 10019708 (hepatic steatosis) |
| | MedDRA PT code 10001627 (alcoholic liver disease) |
| Patient with concurrent | Patient with a check for hepatic steatosis in the column of concurrent illness |
| hepatic steatosis | in the CRF or concurrent illness corresponding to MedDRA PT code |
| | 10019708 (hepatic steatosis) described in the column of other disease: name |
| | of disease |
| Patient with concurrent | Patient with a check for alcoholic hepatopathy in the column of concurrent |
| alcoholic hepatopathy | illness in the CRF or concurrent illness corresponding to MedDRA PT code |
| | 10001627 (alcoholic liver disease) described in the column of other disease: |
| | name of disease |
| Patient with concurrent | Patient with concurrent hepatic impairment who is not a patient with |
| hepatic impairment (other) | concurrent hepatic steatosis or alcoholic hepatopathy |
| Patient with concurrent | Patient with PT corresponding to SMQ code 20000060 (cerebrovascular |
| cerebrovascular disorder | disorders SMQ [scope: narrow]) described in the column of concurrent |

| Term | Definition |
|---|---|
| | illness: other disease: name of disease or medical history in the CRF |
| Age | If the month and day of starting treatment is smaller than the month and day |
| | of birth, age will be calculated as year of starting treatment - year of birth - 1. |
| | If the month and day of starting treatment is equal to or greater than the |
| | month and day of birth, age will be calculated as year of starting treatment - |
| | year of birth. |
| | If the month and day of birth is unknown, January 1 will be used for |
| | calculation. If the day of birth is unknown, 1 will be used for calculation. |
| Young, middle-aged, or | Patient aged 15 years or older and 74 years or younger |
| young-old patient | |
| Old-old patient | Patient aged 75 years or older |
| BMI | BMI will be calculated as body weight (kg) / [0.0001 × height (cm) × height |
| | (cm)]. BMI will be displayed to one decimal place by rounding. |
| Concomitant drug (at the | Concomitant drug that is started before the start of treatment with Zacras and |
| start of treatment with | is not terminated on the day before the start of treatment with Zacras, or |
| Zacras) | concomitant drug that is started on the start day of treatment with Zacras |
| Concomitant drug (during | Concomitant drug used during a period from the start day of treatment with |
| the survey period) | Zacras to the end day of treatment with Zacras |
| Concomitant drug (at the end | Concomitant drug used on the end day of treatment with Zacras |
| of treatment with Zacras) | |
| Antihypertensive used | Drug described in the column for details on the use of other antihypertensive |
| within 2 months before the | in the CRF that is started before the start day of treatment with Zacras and |
| start of treatment with | used within 2 months (60 days) before the start of treatment with Zacras |
| Zacras | (excluding drugs that are started on the start day of treatment with Zacras) |
| Antidiabetic | Drugs with a NHI drug code starting with 396, 2492, or 249941 |
| Antidyslipidemic | Drugs with a NHI drug code starting with 218 or any of the following 7-digit |
| | numbers: |
| | 2190101, 2190102, 2190103, 2190104 |
| Antihyperuricemic | Drugs with a NHI drug code starting with 394 |
| Antihypertensive | ACE inhibitors, angiotensin receptor blockers (ARBs), diuretics (thiazide |
| | and thiazide analogue diuretics), calcium antagonists (hereinafter referred to |
| | as Ca antagonists), direct renin inhibitors, aldosterone |
| | antagonists/potassium-sparing diuretics, vasodilators, β-blockers, central |
| | sympathetic inhibitors, $\alpha\beta$ -blockers, $\alpha_1$ -blockers, fixed-dose combination: |
| | ARB + diuretic, fixed-dose combination: ARB + Ca antagonist, fixed-dose |

| Term | Definition |
|---|---|
| | combination: Ca antagonist + statin, and fixed-dose combination: ARB + Ca |
| | antagonist + diuretic in a list of antihypertensives in the Guidelines for the |
| | Management of Hypertension 2014 (JSH2014) |
| ACE inhibitor | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with the |
| | following 4-digit number: |
| | 2144 |
| | Generic name: captopril, enalapril maleate, perindopril erbumine, lisinopril |
| | hydrate, alacepril, delapril hydrochloride, benazepril hydrochloride, |
| | cilazapril hydrate, imidapril hydrochloride, temocapril hydrochloride, |
| | quinapril hydrochloride, trandolapril |
| ARB | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2149039, 2149040, 2149041, 2149042, 2149044, 2149046, 2149048, |
| | 2149110, 2149111, 2149112, 2149113, 2149119, 2149116, 2149114, |
| | 2149117, 2149118, 2149115, 2149120, 2149122 |
| | Generic name: losartan potassium, candesartan cilexetil, valsartan, |
| | telmisartan, olmesartan medoxomil, irbesartan, azilsartan, losartan |
| | potassium/hydrochlorothiazide, candesartan cilexetil/hydrochlorothiazide, |
| | valsartan/hydrochlorothiazide, telmisartan/hydrochlorothiazide, |
| | irbesartan/trichlormethiazide, candesartan cilexetil/amlodipine besilate, |
| | valsartan/amlodipine besilate, telmisartan/amlodipine besilate, |
| | irbesartan/amlodipine besilate, olmesartan medoxomil/azelnidipine, |
| | valsartan/cilnidipine, azilsartan/amlodipine besilate, telmisartan/amlodipine |
| | besilate/hydrochlorothiazide |
| Diuretic (thiazide and | Drugs described in the column for details on the use of other |
| thiazide analogue diuretic) | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2132003, 2132004, 2132006, 2149103, 2149012, 2135001, 2149007, |
| | 2149003, 2149110, 2149111, 2149112, 2149113, 2149119, 2149122 |
| | Generic name: trichlormethiazide, hydrochlorothiazide, |
| | benzylhydrochlorothiazide, indapamide, mefruside, tripamide, meticrane, |
| | losartan potassium/hydrochlorothiazide, candesartan |
| | cilexetil/hydrochlorothiazide, valsartan/hydrochlorothiazide, |
| | telmisartan/hydrochlorothiazide, irbesartan/trichlormethiazide, |
| | telmisartan/amlodipine besilate/hydrochlorothiazide |

| Term | Definition |
|---|---|
| HCTZ | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2132004, 2149110, 2149111, 2149112, 2149113, 2149122 |
| | Generic name: hydrochlorothiazide, losartan potassium/hydrochlorothiazide, |
| | candesartan cilexetil/hydrochlorothiazide, valsartan/hydrochlorothiazide, |
| | telmisartan/hydrochlorothiazide, telmisartan/amlodipine |
| | besilate/hydrochlorothiazide |
| Dose of HCTZ | The dose of HCTZ is the maximum dose in patients receiving HCTZ. |
| Ca antagonist | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2171022, 2171014, 2171019, 2171020, 2149019, 2149022, 2149043, |
| | 2149027, 2149034, 2149037, 2149038, 2171021, 2149035, 2149030, |
| | 2171006, 2149116, 2149114, 2149117, 2149118, 2149115, 2190101, |
| | 2190102, 2190103, 2190104, 2149120, 2149122 |
| | Generic name: amlodipine besilate, nifedipine, nisoldipine, nitrendipine, |
| | nicardipine hydrochloride, nilvadipine, azelnidipine, manidipine |
| | hydrochloride, efonidipine hydrochloride ethanol, cilnidipine, aranidipine, |
| | benidipine hydrochloride, felodipine, barnidipine hydrochloride, diltiazem |
| | hydrochloride, candesartan cilexetil/amlodipine besilate, |
| | valsartan/amlodipine besilate, telmisartan/amlodipine besilate, |
| | irbesartan/amlodipine besilate, olmesartan medoxomil/azelnidipine, |
| | amlodipine besilate/atorvastatin calcium hydrate, valsartan/cilnidipine, |
| | telmisartan/amlodipine besilate/hydrochlorothiazide |
| Direct renin inhibitor | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with the |
| | following 7-digit number: |
| | 2149047 |
| | Generic name: aliskiren fumarate |
| Aldosterone | Drugs described in the column for details on the use of other |
| antagonist/potassium-sparing | antihypertensive in the CRF that have a NHI drug code starting with any of |
| diuretic | the following 7-digit numbers: |
| | 2133001, 2149045, 2133002 |
| | Generic name: spironolactone, eplerenone, triamterene |
| Aldosterone antagonist | Drugs described in the column for details on the use of other |

| Term | Definition |
|---|---|
| | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2133001, 2149045, |
| | Generic name: spironolactone, eplerenone |
| Potassium-sparing diuretic | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with the |
| | following 7-digit number: |
| | 2133002 |
| | Generic name: triamterene |
| Diuretic | Diuretics (thiazide and thiazide analogue diuretics) or potassium-sparing |
| | diuretics described in the column for details on the use of other |
| | antihypertensive in the CRF |
| Vasodilator | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with the |
| | following 7-digit number: |
| | 2142004 |
| | Generic name: hydralazine hydrochloride |
| β-blocker | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2123011, 2123016, 2149700, 2149031, 2149010, 2123001, 2149029, |
| | 2123008, 2149014, 2149021, 2149028, 2123015, 2123005, 2149025, |
| | 2123009, 2149011 |
| | Generic name: atenolol, bisoprolol fumarate, bisoprolol, betaxolol |
| | hydrochloride, metoprolol tartrate, acebutolol hydrochloride, celiprolol |
| | hydrochloride, propranolol hydrochloride, nipradilol, tilisolol hydrochloride, |
| | nadolol, carteolol hydrochloride, pindolol |
| Central sympathetic inhibitor | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2149001, 2149017, 2145001 |
| | Generic name: clonidine hydrochloride, guanabenz acetate, methyldopa |
| | hydrate |
| αβ-blocker | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |

| Term | Definition |
|---|---|
| | 2149032, 2149018, 2123014, 2149009, 2149036 |
| | Generic name: carvedilol, amosulalol hydrochloride, arotinolol |
| | hydrochloride, labetalol hydrochloride, bevantolol hydrochloride |
| α <sub>1</sub> -blocker | Drugs described in the column for details on the use of other |
| | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2149026, 2149015, 2149023, 2149002, 2149020 |
| | Generic name: doxazosin mesilate, bunazosin hydrochloride, terazosin |
| | hydrochloride hydrate, prazosin hydrochloride, urapidil |
| Fixed-dose combination: | Drugs described in the column for details on the use of other |
| ARB + diuretic | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2149110, 2149111, 2149112, 2149113, 2149119, 2149122 |
| | Generic name: losartan potassium/hydrochlorothiazide, candesartan |
| | cilexetil/hydrochlorothiazide, valsartan/hydrochlorothiazide, |
| | telmisartan/hydrochlorothiazide, irbesartan/trichlormethiazide, |
| | telmisartan/amlodipine besilate/hydrochlorothiazide |
| Fixed-dose combination: | Drugs described in the column for details on the use of other |
| ARB + Ca antagonist | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2149116, 2149114, 2149117, 2149118, 2149115, 2149120, 2149122 |
| | Generic name: candesartan cilexetil/amlodipine besilate, |
| | valsartan/amlodipine besilate, telmisartan/amlodipine besilate, |
| | irbesartan/amlodipine besilate, olmesartan medoxomil/azelnidipine, |
| | valsartan/cilnidipine, telmisartan/amlodipine besilate/hydrochlorothiazide |
| Fixed-dose combination: | Drugs described in the column for details on the use of other |
| ARB + Ca antagonist + | antihypertensive in the CRF that have a NHI drug code starting with the |
| diuretic | following 7-digit number: |
| | 2149122 |
| | Generic name: telmisartan/amlodipine besilate/hydrochlorothiazide |
| Fixed-dose combination: Ca | Drugs described in the column for details on the use of other |
| antagonist + statin | antihypertensive in the CRF that have a NHI drug code starting with any of |
| | the following 7-digit numbers: |
| | 2190101, 2190102, 2190103, 2190104 |
| | Generic name: amlodipine besilate/atorvastatin calcium hydrate |
| Other (antihypertensive) | Vasodilators, $\beta\text{-blockers},$ central sympathetic inhibitors, $\alpha\beta\text{-blockers},$ and |

| Term | Definition |
|---|---|
| | $\alpha_1$ -blockers described in the column for details on the use of other |
| | antihypertensive in the CRF |
| Number of concomitant | The number of drugs described in the column for details on the use of other |
| drugs (antihypertensive other | antihypertensive in the CRF will be tabulated. The fixed-dose combination |
| than Zacras) | will be tabulated as one drug. For instance, "fixed-dose combination: ARB + |
| | diuretic" used concomitantly will be tabulated as one drug. |
| eGFR (mL/min/1.73 m <sup>2</sup> ) | eGFR will be calculated as 194 $\times$ serum creatinine [mg/dL] <sup>-1.094</sup> $\times$ age |
| | [years] <sup>-0.287</sup> (× 0.739 for females). eGFR will be displayed as an integer by |
| | rounding. |
| Summary statistics | Number of patients, mean, standard deviation, minimum, first quartile, |
| | median, third quartile, maximum |

# 1.2 Number of Digits to be Displayed

| Term | Definition |
|---|---|
| Percentage (%) | Incidence of AE or ADR, etc.: |
| | Displayed to two decimal places by rounding |
| | Other: |
| | Displayed to one decimal place by rounding |
| Summary statistics | Mean, median, first quartile, and third quartile: |
| | Displayed to one lower digit than raw data by rounding |
| | Standard deviation: |
| | Displayed to two lower digits than raw data by rounding |
| | Minimum and maximum: |
| | Displayed to the same number of digits as raw data |
| P-value | P-value will be displayed to three decimal places by rounding down. |
| | P-value rounded down to less than 0.001 will be displayed as p<0.001. |

# 1.3 Level of Significance, Confidence Coefficient

Level of significance: 5% (two-sided test)

Confidence coefficient: 95% (two-sided estimate)

# 1.4 Handling of Test/Measurement Data

Test/measurement data will be handled in accordance with the criteria described below (with 1 month as 30 days). If there are multiple pieces of data at the same specified time point, data on the test day closest to the specified day of assessment will be employed, and the latest data among different pieces of data on different days with the same deviation from the specified day of assessment will be

employed. At the final assessment\*, values measured on the day closest to the start date of treatment with Zacras + 375 days will be employed. Values measured 16 days or more after the end day of treatment with Zacras will not be employed.

The number of days from the start day of treatment with Zacras is 1 day for the start day of treatment with Zacras and -1 day for the previous day.

\* After 12 months of treatment with Zacras (or at discontinuation of treatment with Zacras)

| Time point of test | Permissible range (number of days from the start day of treatment) | Specified day of assessment |
|---|---|---|
| At the start of treatment | -90 to -1 | Start date of treatment |
| After 1 month of treatment | 2 to 45 | Start date of treatment + 30 |
| After 2 months of treatment | 46 to 75 | Start date of treatment + 60 |
| After 3 months of treatment | 76 to 105 | Start date of treatment + 90 |
| After 4 months of treatment | 106 to 135 | Start date of treatment + 120 |
| After 5 months of treatment | 136 to 165 | Start date of treatment + 150 |
| After 6 months of treatment | 166 to 195 | Start date of treatment + 180 |
| After 7 months of treatment | 196 to 225 | Start date of treatment + 210 |
| After 8 months of treatment | 226 to 255 | Start date of treatment + 240 |
| After 9 months of treatment | 256 to 285 | Start date of treatment + 270 |
| After 10 months of treatment | 286 to 315 | Start date of treatment + 300 |
| After 11 months of treatment | 316 to 345 | Start date of treatment + 330 |
| After 12 months of treatment | 346 to 375 | Start date of treatment + 360 |
| At the final assessment | 1 to 375 | Start date of treatment + 375 |

### 2.0 Disposition of Patients (Patient Composition Diagram)

(1) Patients included in tabulation/analysis

Enrolled patients

### (2) Data tabulated/analyzed

The number of enrolled patients, number of medical institutions involved in patient registration, number of patients from whom the CRF is collected, number of patients from whom the CRF is not collected, number of finalized patients, number of non-finalized patients, number of patients included in safety evaluation, number of patients excluded from safety evaluation, number of patients included in efficacy evaluation, and number of patients excluded from efficacy evaluation will be tabulated.

For the number of medical institutions involved in patient registration, one medical institution with different departments should not be counted more than once.

For patients from whom the CRF is not collected, the number of patients by reason for failure to collect will be tabulated.

For patients excluded from safety evaluation and those excluded from efficacy evaluation, the number of patients by reason for exclusion will be tabulated, and excluded patients will be listed

Patients meeting any of the criteria listed below will be handled as described below regarding whether to employ them or not.

| Criterion | Safety<br>evaluation | Efficacy evaluation |
|---|---|---|
| Prescription before the contract period | × | × |
| [posterior finding] | | |
| Registration 15 days or more after | × | × |
| prescription of Zacras [posterior finding] | | |
| Non-target disease | 0 | × |
| Deviation from exclusion criteria | 0 | × |
| Failure to confirm the intake of Zacras [after | × | × |
| the patient enrollment period] | | |
| Unavailability of follow-up CRF | 0 | 0 |
| It is unknown whether the patient experienced | × | × |
| an AE | | |

o: employed, x: excluded or not employed

### (3) Table/figure number

Figure 2.0-1, Table 2.0-1

### 3.0 Patient Demographics and Baseline Characteristics

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

### (2) Data tabulated/analyzed

For each variable, patients will be categorized as described below, and the number and proportion of patients will be tabulated.

Variable Category Sex Male, female Summary statistics Age <65 years, ≥65 years <65 years, 65 to <75 years,  $\ge 75$  years Duration of disease <1 year, 1 to <3 years, 3 to <5 years,  $\geq$ 5 years, unknown Diagnostic category (at the start of Outpatient, inpatient treatment with Zacras) Predisposition to No, yes, unknown hypersensitivity Concurrent illness No, yes Diabetes, dyslipidemia, hyperuricemia, cardiac failure, coronary artery disease (myocardial infarction (including old myocardial infarction), Disposition angina, or other), atrial fibrillation, renal impairment (chronic kidney (multiple disease (CKD) [diabetic nephropathy, nephrosclerosis, or other] or tabulation) other), hepatic impairment (hepatic steatosis, alcoholic hepatopathy, or other), cerebrovascular disorder Medical history No, yes, unknown Body weight (kg) Summary statistics  $<40, 40 \text{ to } <50, 50 \text{ to } <60, 60 \text{ to } <70, \ge 70, \text{ not measured}$ BMI  $(kg/m^2)$ Summary statistics <18.5, 18.5 to <25.0, 25.0 to <30.0,  $\ge30.0$ , unknown eGFR [at the start of Summary statistics treatment] <15, 15 to <30, 30 to <45, 45 to <60, 60 to <90, ≥90, unknown  $(mL/min/1.73 m^2)$ Smoking history Never smoked, current smoker, past smoker, unknown Drinking history (drink alcoholic Yes, no, unknown beverage almost every day)

| Presence or absence | |
|------------------------|---------|
| of breast-feeding (at | |
| the start of treatment | No, yes |
| with Zacras) [only | |
| females] | |

Table 3.0-1

# 4.0 Treatment Given

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

# (2) Data tabulated/analyzed

For each variable, patients will be categorized as described below, and the number and proportion of patients will be tabulated.

| Variable Variable | Category |
|---|---|
| Initial dose of Zacras | LD, HD |
| Presence or absence | |
| of change in daily | No, yes |
| dose of Zacras | |
| | $LD{\rightarrow}HD, HD{\rightarrow}LD, LD{\rightarrow}HD{\rightarrow}LD, HD{\rightarrow}LD{\rightarrow}HD$ |
| Disposition | * This categorization is an example and subject to change depending on |
| | actual data. |
| Duration of treatment | 1 to 180 days, 181 to 360 days, ≥361 days |
| with Zacras | 1 to 100 days, 101 to 300 days, ≥301 days |
| Presence or absence | |
| of discontinuation of | No, yes |
| treatment with Zacras | |
| Reason for | Successful achievement of treatment goal, AE, patient's failure to visit |
| discontinuation of | the hospital such as transfer to another hospital, insufficient efficacy, |
| treatment with Zacras | other |
| Azilsartan and | Azilsartan 20 mg, amlodipine 2.5 mg, amlodipine 5 mg, combined use |
| amlodipine used | of azilsartan 20 mg/amlodipine 2.5 mg, combined use of azilsartan |
| before the start of | 20 mg/amlodipine 5 mg, other |
| treatment with Zacras | 20 11.9 41.110 41.19.10 11.19. |
| Switching to Zacras | Azilsartan 20 mg→Zacras LD, azilsartan 20 mg→Zacras HD, |
| (by ingredient/dose) | amlodipine 2.5 mg→Zacras LD, amlodipine 5 mg→Zacras HD, |
| | combined use of azilsartan 20 mg/amlodipine 2.5 mg→Zacras LD, |
| | combined use of azilsartan 20 mg/amlodipine 5 mg→Zacras HD, other |
| Switching to Zacras | Azilsartan→Zacras, amlodipine→Zacras, combined use of |
| (by ingredient) | azilsartan/amlodipine→Zacras, other |
| Treatment with | |
| antihypertensive other | |
| than Zacras (at the | No, yes |
| start of treatment with | |
| Zacras) | |

| <b></b> | |
|---|---|
| Disposition (multiple tabulation)* Antihypertensive other than Zacras: treatment with HCTZ (at the start of treatment with Zacras) | ACE inhibitor, ARB, diuretic (thiazide and thiazide analogue diuretic), Ca antagonist, direct renin inhibitor, aldosterone antagonist, potassium-sparing diuretic, fixed-dose combination: ARB + diuretic, fixed-dose combination: ARB + Ca antagonist, fixed-dose combination: ARB + Ca antagonist + diuretic, fixed-dose combination: Ca antagonist + statin, other |
| Disposition | 6.25 mg, 12.5 mg, other |
| Treatment with antihypertensive other than Zacras (during the survey period) | No, yes |
| Disposition (multiple tabulation)* | ACE inhibitor, ARB, diuretic (thiazide and thiazide analogue diuretic), Ca antagonist, direct renin inhibitor, aldosterone antagonist, potassium-sparing diuretic, fixed-dose combination: ARB + diuretic, fixed-dose combination: ARB + Ca antagonist, fixed-dose combination: ARB + Ca antagonist + diuretic, fixed-dose combination: Ca antagonist + statin, other |
| Antihypertensive other than Zacras: treatment with HCTZ (during the survey period) | No, yes |
| Disposition | 6.25 mg, 12.5 mg, other |
| Treatment with antihypertensive other than Zacras (within 2 months before the start of treatment with Zacras) | No, yes |
| Disposition (multiple tabulation)* | ACE inhibitor, ARB, diuretic (thiazide and thiazide analogue diuretic), Ca antagonist, direct renin inhibitor, aldosterone antagonist, potassium-sparing diuretic, fixed-dose combination: ARB + diuretic, |

| | fixed-dose combination: ARB + Ca antagonist, fixed-dose combination: ARB + Ca antagonist + diuretic, fixed-dose combination: Ca antagonist |
|---|---|
| | + statin, other |
| Number of | |
| concomitant drugs | |
| (antihypertensive | |
| other than Zacras) | |
| (at the start of treatment with Zacras) | $0, 1, 2, 3, 4, 5, \ge 6$ |
| (at the end of treatment with Zacras) | $0, 1, 2, 3, 4, 5, \ge 6$ |
| Concomitant non-antihypertensive drug (during the survey period) | No, yes |
| Disposition (multiple tabulation) | Antidiabetic, antidyslipidemic, antihyperuricemic, other |

<sup>\*</sup> For fixed-dose combinations, individual ingredients will be tabulated separately. If "fixed-dose combination: ARB + diuretic" is used concomitantly, for instance, "ARB" and "diuretic" will also be tabulated.

Table 4.0-1

# 5.0 Tabulation/Analysis of Safety

# 5.1 Occurrence of Adverse Events and Adverse Drug Reactions/Infections

### 5.1.1 Occurrence of Adverse Events

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with an AE | Number of patients who experienced an AE |
| Number of AE | Number of reported AE. Multiple episodes of the same AE (PT) in the same patient will be tabulated as the total number of episodes. |
| Incidence of AE | The incidence of AE will be calculated as number of patients with an AE/number of patients included in safety evaluation $\times$ 100. |
| Type of AE | AEs will be classified by SOC and then tabulated by PT. For laboratory tests, AEs will be classified by SOC, then sorted by HLGT, and finally tabulated by PT. For SOC, the number of patients with an AE and the incidence of AE will be listed by SOC internationally agreed order. For PT, the number of patients with an AE and the incidence of AE will be listed in ascending order of PT code. Multiple episodes of the same AE (PT) in the same patient will be tabulated as 1 patient. |

# (3) Table/figure number

Table 5.1-1

# 5.1.2 Occurrence of Adverse Drug Reactions/Infections

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with | Number of patients who experienced an ADR, etc. |
| an ADR, etc. | realised of patients who experienced an ADR, etc. |
| | Number of reported ADR, etc. Multiple episodes of the same ADR, |
| Number of ADR, etc. | etc. (PT) in the same patient will be tabulated as the total number of |
| | episodes. |
| Incidence of ADR, etc. | The incidence of ADR, etc. will be calculated as number of patients |

| | with an ADR, etc./number of patients included in safety evaluation |
|---|---|
| | × 100. |
| | ADRs, etc. will be classified by SOC and then tabulated by PT. For |
| | laboratory tests, ADRs, etc. will be classified by SOC, then sorted |
| | by HLGT, and finally tabulated by PT. |
| Type of ADR, etc. | For SOC, the number of patients with an ADR, etc. and the |
| | incidence of ADR, etc. will be listed by SOC internationally agreed |
| | order. |
| | For PT, the number of patients with ADR, etc. and the incidence of |
| | ADR, etc. will be listed in ascending order of PT code. Multiple |
| | episodes of the same ADR, etc. (PT) in the same patient will be |
| | tabulated as 1 patient. |

Table 5.1-2

- 5.2 Occurrence of Adverse Events and Adverse Drug Reactions/Infections in Patients Excluded from Safety Evaluation
  - 5.2.1 Occurrence of Adverse Events
    - (1) Patients included in tabulation/analysis
      - Patients excluded from safety evaluation
    - (2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with an AE | Number of patients who experienced an AE |
| Number of AE | Number of reported AE. Multiple episodes of the same AE (PT) in the same patient will be tabulated as the total number of episodes. |
| Incidence of AE | The incidence of AE will be calculated as number of patients with an AE/number of patients excluded from safety evaluation × 100. |
| Type of AE | AEs will be classified by SOC and then tabulated by PT. For laboratory tests, AEs will be classified by SOC, then sorted by HLGT, and finally tabulated by PT. For SOC, the number of patients with an AE and the incidence of AE will be listed by SOC internationally agreed order. For PT, the number of patients with an AE and the incidence of AE will be listed in ascending order of PT code. Multiple episodes of the same AE (PT) in the same patient will be tabulated as 1 patient. |

(3) Table/figure number
Table 5.2-1

# 5.2.2 Occurrence of Adverse Drug Reactions/Infections

(1) Patients included in tabulation/analysis

Patients excluded from safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with an ADR, etc. | Number of patients who experienced an ADR, etc. |
| Number of ADR, etc. | Number of reported ADR, etc. Multiple episodes of the same ADR, etc. (PT) in the same patient will be tabulated as the total number of episodes. |
| Incidence of ADR, etc. | The incidence of ADR, etc. will be calculated as number of patients with an ADR, etc./number of patients excluded from safety evaluation × 100. |
| Type of ADR, etc. | ADRs, etc. will be classified by SOC and then tabulated by PT. For laboratory tests, ADRs, etc. will be classified by SOC, then sorted by HLGT, and finally tabulated by PT. For SOC, the number of patients with an ADR, etc. and the incidence of ADR, etc. will be listed by SOC internationally agreed order. For PT, the number of patients with ADR, etc. and the incidence of ADR, etc. will be listed in ascending order of PT code. Multiple episodes of the same ADR, etc. (PT) in the same patient will be tabulated as 1 patient. |

(3) Table/figure number

Table 5.2-2

- 5.3 Occurrence of Adverse Events and Adverse Drug Reactions/Infections by Seriousness, Time of Onset, and Outcome
  - 5.3.1 Occurrence of Adverse Events by Seriousness, Time of Onset, and Outcome
    - (1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

AEs will be categorized for each variable as described below, and the type of AE will be tabulated.

| Variable | Category |
|---|---|
| Seriousness | Serious, non-serious |
| Time of onset | Days 1 to 180, Days 181 to 360, Day 361 or later |
| Outcome | Recovered, recovering, not recovered, recovered with sequelae, fatal, unknown |

The type of AE will be tabulated as described below.

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients | Number of patients who experienced an AE by SOC/PT |
| Number of AE | Number of reported AE by SOC/PT |
| | AEs will be classified by SOC and then tabulated by PT. For |
| | laboratory tests, AEs will be classified by SOC, then sorted by |
| Type of AE | HLGT, and finally tabulated by PT. |
| | AEs will be listed for SOC by SOC internationally agreed order and |
| | for PT in ascending order of PT code. |
| | Multiple episodes of the same AE (PT) in the same patient will be |
| | tabulated by category as the total number of episodes (for instance, |
| | one episode of serious diarrhoea and one episode of non-serious |
| | diarrhoea in the same patient will be counted once in the respective |
| | categories). |

# (3) Table/figure number

Table 5.3-1

# 5.3.2 Occurrence of Adverse Drug Reactions/Infections by Seriousness, Time of Onset, and Outcome

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

# (2) Data tabulated/analyzed

ADRs, etc. will be categorized for each variable as described below, and the type of ADR will be tabulated.

| Variable | Category |
|---|---|
| Seriousness | Serious, non-serious |
| Time of onset | Days 1 to 180, Days 181 to 360, Day 361 or later |
| Outcome | Recovered, recovering, not recovered, recovered with sequelae, fatal, unknown |

The type of ADR, etc. will be tabulated as described below.

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients | Number of patients who experienced an ADR, etc. by SOC/PT |
| Number of ADR, etc. | Number of reported ADR, etc. by SOC/PT |
| | ADRs, etc. will be classified by SOC and then tabulated by PT. For |
| Type of ADR, etc. | laboratory tests, ADRs, etc. will be classified by SOC, then sorted |
| | by HLGT, and finally tabulated by PT. |
| | ADRs, etc. will be listed for SOC by SOC internationally agreed |
| | order and for PT in ascending order of PT code. |
| | Multiple episodes of the same ADR, etc. (PT) in the same patient |
| | will be tabulated by category as the total number of episodes (for |
| | instance, one episode of serious diarrhoea and one episode of |
| | non-serious diarrhoea in the same patient will be counted once in |
| | the respective categories). |

# (3) Table/figure number

Table 5.3-2

- 5.4 Incidence of Adverse Drug Reaction/Infection by Factors Related to Patient Demographics and Baseline Characteristics and Treatment Given
  - (1) Patients included in tabulation/analysis

    Patients included in safety evaluation

# (2) Data tabulated/analyzed

ADRs, etc. will be categorized for each variable as described below, and the incidence of ADR, etc. will be tabulated.

ADRs, etc. will be categorized for each variable as described below, and the type of ADR, etc. will be tabulated. The type of ADR, etc. will be tabulated as described in Section 5.1. For disposition of treatment with antihypertensive other than Zacras (at the start of treatment with Zacras) and disposition of treatment with antihypertensive other than Zacras (during the survey period), "other" will not be tabulated.

| Variable | Category |
|---|---|
| Sex | Male, female |
| Age | <65 years, ≥65 years |
| | <65 years, 65 to <75 years, ≥75 years |
| Predisposition to | No, yes, unknown |
| hypersensitivity | ivo, yes, unknown |
| Concurrent illness | No, yes |
| | Diabetes, dyslipidemia, hyperuricemia, cardiac failure, coronary |
| Disposition | artery disease, atrial fibrillation, renal impairment, hepatic |
| | impairment, cerebrovascular disorder |
| Initial dose of Zacras | LD, HD |
| Presence or absence | |
| of change in daily | No, yes |
| dose of Zacras | |
| Switching to Zacras | Azilsartan→Zacras, amlodipine→Zacras, combined use of |
| (by ingredient) | azilsartan/amlodipine→Zacras, other |
| Treatment with | |
| antihypertensive other | |
| than Zacras (at the | No, yes |
| start of treatment with | |
| Zacras) | |
| Disposition (multiple | ACE inhibitor ADD diversity Counterconist other |
| tabulation)* | ACE inhibitor, ARB, diuretic, Ca antagonist, other |
| Treatment with | No, yes |

| antihypertensive other | |
|------------------------|----------------------------------------------------|
| than Zacras (during | |
| the survey period) | |
| Disposition | ACE inhibitor, ARB, diuretic, Ca antagonist, other |
| (multiple tabulation)* | |

<sup>\*</sup> For fixed-dose combinations, individual ingredients will be tabulated separately. If "fixed-dose combination: ARB + diuretic" is used concomitantly, for instance, "ARB" and "diuretic" will also be tabulated.

Tables 5.4.2-1 to -26

# 5.5 Listing of Occurrence of Serious Adverse Events and Serious Adverse Drug Reactions/Infections

# 5.5.1 Occurrence of Serious Adverse Events

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with a SAE | Number of patients who experienced a SAE |
| | Number of reported SAE |
| Number of SAE | Multiple episodes of the same SAE (PT) in the same patient will be |
| | tabulated as the total number of episodes. |
| Incidence of SAE | The incidence of SAE will be calculated as number of patients with |
| medence of SAE | a SAE/number of patients included in safety evaluation $\times$ 100. |
| | SAEs will be classified by SOC and then tabulated by PT. For |
| | laboratory tests, SAEs will be classified by SOC, then sorted by |
| | HLGT, and finally tabulated by PT. |
| | For SOC, the number of patients with a SAE and the incidence of |
| Type of SAE | SAE will be listed by SOC internationally agreed order. |
| | For PT, the number of patients with a SAE and the incidence of |
| | SAE will be listed in ascending order of PT code. |
| | Multiple episodes of the same SAE (PT) in the same patient will be |
| | tabulated as 1 patient. |
| | The number of patients with a SAE not related to Zacras will be |
| | presented in parentheses. |

# (3) Table/figure number

Table 5.5-1

# 5.5.2 Occurrence of Serious Adverse Drug Reactions/Infections

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with | Number of patients who experienced a serious ADR, etc. |
| a serious ADR, etc. | |
| Number of serious ADR, | Number of reported serious ADR, etc. |

| etc. | Multiple episodes of the same serious ADR, etc. (PT) in the same |
|---|---|
| | patient will be tabulated as the total number of episodes. |
| Incidence of serious ADR, etc. | The incidence of serious ADR, etc. will be calculated as number of patients with a serious ADR, etc./number of patients included in safety evaluation $\times$ 100. |
| Type of serious ADR, etc. | Serious ADRs, etc. will be classified by SOC and then tabulated by PT. For laboratory tests, serious ADRs, etc. will be classified by SOC, then sorted by HLGT, and finally tabulated by PT. For SOC, the number of patients with a serious ADR, etc. and the incidence of serious ADR, etc. will be listed by SOC internationally agreed order. For PT, the number of patients with a serious ADR, etc. and the incidence of serious ADR, etc. will be listed in ascending order of PT code. |

Table 5.5-2

- 5.6 Listing of Occurrence of Serious Adverse Events and Serious Adverse Drug Reactions/Infections in Patients Excluded from Safety Evaluation
  - 5.6.1 Occurrence of Serious Adverse Events
    - (1) Patients included in tabulation/analysis

Patients excluded from safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with a SAE | Number of patients who experienced a SAE |
| Number of SAE | Number of reported SAE |
| | Multiple episodes of the same SAE (PT) in the same patient will |
| | be tabulated as the total number of episodes. |
| Incidence of SAE | The incidence of SAE will be calculated as number of patients |
| | with a SAE/number of patients included in safety evaluation × |
| | 100. |
| Type of SAE | SAEs will be classified by SOC and then tabulated by PT. For |
| | laboratory tests, SAEs will be classified by SOC, then sorted by |
| | HLGT, and finally tabulated by PT. |
| | For SOC, the number of patients with a SAE and the incidence of |

| SAE will be listed by SOC internationally agreed order. |
|-----------------------------------------------------------------|
| For PT, the number of patients with a SAE and the incidence of |
| SAE will be listed in ascending order of PT code. |
| Multiple episodes of the same SAE (PT) in the same patient will |
| be tabulated as 1 patient. |
| The number of patients with a SAE not related to Zacras will be |
| presented in parentheses. |

Table 5.6-1

# 5.6.2 Occurrence of Serious Adverse Drug Reactions/Infections

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with a serious ADR, etc. | Number of patients who experienced a serious ADR, etc. |
| Number of serious ADR, etc. | Number of reported serious ADR, etc. Multiple episodes of the same serious ADR, etc. (PT) in the same patient will be tabulated as the total number of episodes. |
| Incidence of serious ADR, etc. | The incidence of serious ADR, etc. will be calculated as number of patients with a serious ADR, etc./number of patients included in safety evaluation × 100. |
| Type of serious ADR, etc. | Serious ADRs, etc. will be classified by SOC and then tabulated by PT. For laboratory tests, serious ADRs, etc. will be classified by SOC, then sorted by HLGT, and finally tabulated by PT. For SOC, the number of patients with a serious ADR, etc. and the incidence of serious ADR, etc. will be listed by SOC internationally agreed order. For PT, the number of patients with a serious ADR, etc. and the incidence of serious ADR, etc. will be listed in ascending order of PT code. |

# (3) Table/figure number

Table 5.6-2

### 5.7 Changes in Test/Measurement Data over Time

### 5.7.1 Vital Signs (Pulse Rate)

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

# (2) Data tabulated/analyzed

Analyses described below will be performed for patients who have relevant data both before and after treatment with Zacras.

For pulse rate (bpm), summary statistics will be calculated for measured values at each time point of measurement [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment]. For the change from the start of treatment with Zacras, summary statistics will be calculated.

# (3) Table/figure number

Table 5.7-1

### 5.7.2 Laboratory Tests

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

### (2) Data tabulated/analyzed

Analyses described below will be performed for patients who have relevant data both before and after treatment with Zacras.

For white blood cell count, platelet count, AST, ALT,  $\gamma$ -GTP, serum creatinine, BUN, and serum potassium, summary statistics will be calculated for test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment]. For the change from the start of treatment with Zacras, summary statistics will be calculated.

### (3) Table/figure number

Table 5.7-2

### 6.0 Tabulation/Analysis of Efficacy

- 6.1 Changes in Blood Pressure over Time
  - (1) Patients included in tabulation/analysis

Patients included in efficacy evaluation

(2) Data tabulated/analyzed

Analyses described below will be performed for patients who have relevant data both before and after treatment with Zacras.

For systolic and diastolic blood pressure, summary statistics and 95% CI for the mean will be calculated for test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment]. The mean and standard deviation of test data will be illustrated.

In addition, the proportion of patients with normal blood pressure at each time point of test will be tabulated. The proportion of patients with normal blood pressure will be illustrated. A patient with normal blood pressure is defined as a patient meeting both criteria listed below. A patient with missing data on systolic and/or diastolic blood pressure will be handled as a patient with missing data.

- •Systolic blood pressure <140 mmHg
- •Diastolic blood pressure <90 mmHg
- (3) Table/figure number

Table 6.1.1, Table 6.1.2, Figure 6.1.1, Figure 6.1.2

- 6.2 Changes in Blood Pressure over Time in Patients Who Switch from the Combined Use of Azilsartan and Amlodipine
  - (1) Patients included in tabulation/analysis

Patients included in efficacy evaluation who switch from combined use

(2) Data tabulated/analyzed

Analyses described below will be performed for patients who have relevant data both before and after treatment with Zacras.

For systolic and diastolic blood pressure, summary statistics and 95% CI for the mean will be calculated for test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment]. For the change from the start of treatment with Zacras, summary statistics and 95% CI for the mean will be calculated. The mean and standard deviation of test data and change will be illustrated. The percentage change from the start of treatment with Zacras ((test data at each time point of test - test data at the start of treatment with Zacras)  $\div$  test data at the start of treatment with Zacras × 100), summary statistics will be calculated. The proportion of patients with normal blood pressure at each time point of test will be tabulated. The proportion of patients with normal blood pressure

will be illustrated.

## (3) Table/figure number

Table 6.2.1, Table 6.2.2, Table 6.2.3, Figure 6.2.1-1, Figure 6.2.1-2, Figure 6.2.3

- 6.3 Changes in Blood Pressure over Time in Patients Except for Those Who Switch from the Combined Use of Azilsartan and Amlodipine
  - (1) Patients included in tabulation/analysis

Patients included in efficacy evaluation except for those who switch from combined use

(2) Data tabulated/analyzed

Analyses described below will be performed for patients who have relevant data both before and after treatment with Zacras.

For systolic and diastolic blood pressure, summary statistics and 95% CI for the mean will be calculated for test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment]. For the change from the start of treatment with Zacras, summary statistics and 95% CI for the mean will be calculated, and the paired t-test will be performed. The mean and standard deviation of test data and change will be illustrated. For the percentage change from the start of treatment with Zacras, summary statistics will be calculated.

The proportion of patients with normal blood pressure at each time point of test will be tabulated. The proportion of patients with normal blood pressure will be illustrated.

(3) Table/figure number

Table 6.3.1, Table 6.3.2, Table 6.3.3, Figure 6.3.1-1, Figure 6.3.1-2, Figure 6.3.3

- 6.4 Factors that May Affect the Efficacy
  - (1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

Analyses described below will be performed for patients who have relevant data both before and after treatment with Zacras.

For test data on systolic and diastolic blood pressure at the final assessment, summary statistics and 95% CI for the mean will be calculated by the variables listed below.

| Variable | Category |
|--------------------|---------------------------------------|
| Sex | Male, female |
| Age | <65 years, ≥65 years |
| | <65 years, 65 to <75 years, ≥75 years |
| Concurrent illness | No, yes |
| Disposition (multiple tabulation) | Diabetes, dyslipidemia, hyperuricemia, cardiac failure, coronary artery disease, atrial fibrillation, renal impairment, hepatic impairment, cerebrovascular disorder |
|---|---|
| Initial dose of Zacras | LD, HD |
| Presence or absence | |
| of change in daily | No, yes |
| dose of Zacras | |
| Treatment with | |
| antihypertensive other | |
| than Zacras (at the | No, yes |
| start of treatment with | |
| Zacras) | |
| Disposition (multiple tabulation)* | ACE inhibitor, ARB, diuretic, Ca antagonist, other |
| Treatment with | |
| antihypertensive other | No, yes |
| than Zacras (during | 110, 300 |
| the survey period) | |
| Disposition (multiple tabulation)* | ACE inhibitor, ARB, diuretic, Ca antagonist, other |

<sup>\*</sup> For fixed-dose combinations, individual ingredients will be tabulated separately. If "fixed-dose combination: ARB + diuretic" is used concomitantly, for instance, "ARB" and "diuretic" will also be tabulated.

Table 6.4.1

# Statistical Analysis Plan Specified Drug-Use Survey ("Long-Term Use Survey") on Zacras Combination Tablets LD & HD

| | Takeda Pharmaceut | ical Company Limited |
|-----|-----------------------|-------------------------|
| | P | PD |
| Cor | ntract Organization f | or Statistical Analysis |
| | Responsible Person | |
| | Responsible Person | |
| | Responsible Person | |
| | Responsible Person | |
| | Responsible Person | |

# Table of Contents

| 1.0 | Definitions of Terms, etc. and Handling of Test/Measurement Data | 4 |
|---|---|---|
| 1.1 | Definitions | 4 |
| 1.2 | Number of Digits to be Displayed | 13 |
| 1.3 | Level of Significance | 14 |
| 1.4 | Handling of Test/Measurement Data | 14 |
| 2.0 | Disposition of Patients (Patient Composition Diagram) | 16 |
| 3.0 | Patient Demographics and Baseline Characteristics | 18 |
| 4.0 | Treatment Given | 20 |
| 5.0 | Tabulation/Analysis of Safety | 23 |
| 5.1 | Occurrence of Adverse Events/Infections and Adverse Drug Reactions/Infections | 23 |
| 5.1 | .1 Occurrence of Adverse Events/Infections | 23 |
| 5.1 | .2 Occurrence of Adverse Drug Reactions/Infections | 23 |
| 5.2 | Occurrence of Adverse Events/Infections and Adverse Drug Reactions/Infections in Patients | S |
| | Excluded from Safety Evaluation | 24 |
| 5.2 | .1 Occurrence of Adverse Events/Infections | 24 |
| 5.2 | 2.2 Occurrence of Adverse Drug Reactions/Infections | 25 |
| 5.3 | Occurrence of Adverse Events/Infections and Adverse Drug Reactions/Infections by Seriousness | , |
| | Time of Onset, and Outcome | 25 |
| 5.3 | .1 Occurrence of Adverse Events/Infections by Seriousness, Time of Onset, and Outcome | 25 |
| 5.3 | 2.2 Occurrence of Adverse Drug Reactions/Infections by Seriousness, Time of Onset, and Outcome | 26 |
| 5.4 | Incidence of Adverse Event/Infection and Adverse Drug Reaction/Infection by Factors Related to | ) |
| | Patient Demographics and Baseline Characteristics and Treatment Given | 27 |
| 5.4 | 1.1 Incidence of Adverse Event/Infection by Factors Related to Patient Demographics and Baseline | |
| | Characteristics and Treatment Given | 27 |
| 5.4 | 2.2 Incidence of Adverse Drug Reaction/Infection by Factors Related to Patient Demographics and | i |
| | Baseline Characteristics and Treatment Given | 29 |
| 5.5 | Occurrence of Adverse Events/Infections and Adverse Drug Reactions/Infections by Age Group | 31 |
| 5.5 | .1 Occurrence of Adverse Events/Infections by Age Group | 31 |
| 5.5 | .2 Occurrence of Adverse Drug Reactions/Infections by Age Group | 32 |
| 5.6 | Occurrence of Adverse Events/Infections and Adverse Drug Reactions/Infections by the Presence of | |
| | Absence of Concurrent Hepatic Impairment | 32 |
| 5.6 | 1.1 Occurrence of Adverse Events/Infections by the Presence or Absence of Concurrent Hepatic | 2 |
| | Impairment | 32 |
| 5.6 | 2.2 Occurrence of Adverse Drug Reactions/Infections by the Presence or Absence of Concurrence | t |
| | Hepatic Impairment | 32 |
| 5.7 | Occurrence of Adverse Events/Infections and Adverse Drug Reactions/Infections by the Presence o | r |
| | Absence of Concurrent Renal Impairment | 32 |
| 5.7 | 7.1 Occurrence of Adverse Events/Infections by the Presence or Absence of Concurrent Rena | 1 |

| | Impairment | 33 |
|---|---|---|
| 5.7. | 2 Occurrence of Adverse Drug Reactions/Infections by the Presence or Absence of Concurrent Rena<br>Impairment | |
| <i>5</i> 0 | • | |
| 5.8 | Occurrence of Adverse Drug Reactions/Infections by the Presence or Absence of Concomitant | |
| 5.0 | Antihypertensive Other than Zacras (during the Survey Period) | |
| 5.9 | Listing of Occurrence of Serious Adverse Events/Infections | |
| 5.10 | Listing of Occurrence of Serious Adverse Events/Infections in Patients Excluded from Safety | |
| | Evaluation | |
| 5.11 | Changes in Test/Measurement Data over Time | |
| | 1.1 Vital Signs (Pulse Rate) | |
| | 1.2 Laboratory Tests | |
| 5.12 | Occurrence of Adverse Drug Reactions/Infections by the Presence or Absence of Concomitant ACE | |
| | Inhibitor (during the Survey Period) | |
| 5.13 | Occurrence of Adverse Drug Reactions/Infections by the Presence or Absence of Concomitant | |
| | Aldosterone Antagonist (during the Survey Period) | 38 |
| 5.14 | Occurrence of Adverse Drug Reactions/Infections by the Presence or Absence of Concomitant Renir | 1 |
| | Inhibitor (during the Survey Period) | 38 |
| 5.15 | Occurrence of Adverse Drug Reactions/Infections by the Presence or Absence of Concomitant | t |
| | Diuretic (during the Survey Period) | 39 |
| 5.16 | Occurrence of Adverse Drug Reactions/Infections by the Presence or Absence of Concomitant | t |
| | HCTZ (during the Survey Period) | 39 |
| 6.0 | Tabulation/Analysis of Efficacy | 40 |
| 6.1 | Changes in Blood Pressure over Time | 40 |
| 6.2 | Changes in Blood Pressure over Time <male></male> | 40 |
| 6.3 | Changes in Blood Pressure over Time <female></female> | 40 |
| 6.4 | Changes in Blood Pressure over Time <<65 Years> | 41 |
| 6.5 | Changes in Blood Pressure over Time <65 to 74 Years> | 41 |
| 6.6 | Changes in Blood Pressure over Time <275 Years> | 41 |
| 6.7 | Changes in Blood Pressure over Time < Presence or Absence of Concurrent Hepatic Impairment | t |
| | (No)> | 41 |
| 6.8 | Changes in Blood Pressure over Time < Presence or Absence of Concurrent Hepatic Impairment | t |
| | (Yes)> | 42 |
| 6.9 | Changes in Blood Pressure over Time < Presence or Absence of Concurrent Renal Impairment (No)> | 42 |
| 6.10 | Changes in Blood Pressure over Time < Presence or Absence of Concurrent Renal Impairment (Yes)> | .42 |
| 6.11 | Changes in Blood Pressure over Time < Concomitant Treatment with Zacras HD/HCTZ 6.25 mg (a) | t |
| | the Start of Treatment with Zacras)> | 43 |
| 6.12 | Changes in Blood Pressure over Time < Concomitant Treatment with Zacras HD/HCTZ 12.5 mg (at | |
| | the Start of Treatment with Zacras)> | |
| 6.13 | Proportion of Patients with Normal Blood Pressure | |
| 6 14 | Factors that May Affect the Efficacy | 44 |

# 1.0 Definitions of Terms, etc. and Handling of Test/Measurement Data

# 1.1 Definitions

| Term | Definition |
|---|---|
| Zacras | Zacras Combination Tablets are abbreviated as Zacras in this document. |
| SOC | System organ class listed in the MedDRA/J |
| HLGT | High level group term listed in the MedDRA/J |
| PT | Preferred term listed in the MedDRA/J |
| LLT | Lowest level term listed in the MedDRA/J |
| Enrolled patient | Patient allowed to be enrolled |
| Patient from whom the CRF is collected | Patient from whom the CRF has been obtained |
| Patient from whom the CRF is not collected | Enrolled patient from whom the CRF has not been collected |
| Finalized patient | Patient from whom the CRF is collected who has the date of CRF completion entered into the PMS system or who requires no information on the CRF |
| | status and has not been excluded from the survey |
| Non-finalized patient | Patient from whom the CRF is collected who has not been finalized |
| Patient included in safety | Finalized patient who is included in safety evaluation |
| evaluation | |
| Patient excluded from safety | Finalized patient who is excluded from safety evaluation |
| evaluation | |
| Patient included in efficacy evaluation | Patient included in safety evaluation who is included in efficacy evaluation |
| Patient excluded from | Patient included in safety evaluation who meets neither (1) nor (2) |
| efficacy evaluation | (1) Office blood pressure (systolic): Test data are available both before and |
| | after <sup>1)</sup> treatment with Zacras. |
| | (2) Office blood pressure (diastolic): Test data are available both before and |
| | after <sup>1)</sup> treatment with Zacras. |
| | 1) Values measured after the end of treatment with Zacras will not be |
| | employed. Values measured during the off-treatment period will be employed. |
| Presence or absence of | "Yes" for patients with a change in daily dose at the final assessment versus |
| change in daily dose of | at the start of treatment with Zacras |
| Zacras | |
| Duration of treatment with Zacras | End date of treatment with Zacras - start date of treatment with Zacras + 1 |
| End date of treatment | End date of the final dose described in the column of the end date of |
| | treatment in the CRF; or start date of treatment + 360 days if the end date of |

| Term | Definition |
|---|---|
| | treatment is not described in the CRF and there is a check for "ongoing at 12 |
| | months after the start of treatment with Zacras." |
| Off-treatment period | The off-treatment period will be allowed until the end date of treatment |
| | before suspension of treatment + 90 days. |
| | If the off-treatment period continues beyond the end date of treatment + 90 |
| | days, the end date of treatment is defined as the end date of treatment before |
| | suspension of treatment. |
| Treatment completer | Patient with a duration of treatment with Zacras of ≥ start date of treatment + |
| | 360 days |
| Treatment non-completer | Patient with a duration of treatment with Zacras of ≤ start date of treatment + |
| | 359 days |
| Reason for discontinuation | If the duration of treatment with Zacras is ≤ start date of treatment + 359 |
| of treatment with Zacras | days, the reason for discontinuation of treatment described in the column of |
| | details on the use of Zacras in the CRF will be employed. |
| | If the duration of treatment with Zacras is ≥ start date of treatment + 360 |
| | days, the patient will be handled as a treatment completer; therefore, the |
| | reason for discontinuation of treatment described in the column of details on |
| | the use of Zacras in the CRF will not be employed. |
| Duration of disease | (Start date of treatment with Zacras - time of diagnosis of hypertension + 1) ÷ |
| | 365.25. For time of diagnosis of hypertension, 1 will be used as the day, and |
| | January 1 will be used if the month is unknown. |
| AE, etc. | Abbreviation of "adverse event/infection" |
| | In this document, "adverse event/infection" is used in titles, and "adverse |
| | event, etc." is used in the text and tables. |
| ADR, etc. | Abbreviation of "adverse drug reaction/infection" |
| | AE, etc. other than those assessed by the investigator to be not related to |
| | Zacras |
| | In this document, "adverse drug reaction/infection" is used in titles, and |
| | "adverse drug reaction, etc." is used in the text and tables. |
| SAE, etc. | Abbreviation of "serious adverse event/infection" |
| | Adverse event assessed by the investigator to be serious |
| | Events included in the MedDRA code list in Takeda Medically Significant AE |
| | List will be handled as serious even if assessed by the investigator to be |
| | non-serious. |
| | In this document, "serious adverse event/infection" is used in titles, and |
| | "serious adverse event, etc." is used in the text and tables. |

| Term | Definition |
|---|---|
| Number of patients with an | Number of patients who experienced an AE, etc. or an ADR, etc. |
| AE, etc. or an ADR, etc. | |
| Number of AE, etc. or ADR, | Number of reported AE, etc. or ADR, etc. |
| etc. | |
| Incidence | [When safety is tabulated in patients included in safety evaluation] |
| | The incidence will be calculated as number of patients with an AE, etc. or |
| | an ADR, etc./number of patients included in safety evaluation × 100. |
| | [When safety is tabulated in patients excluded from safety evaluation] |
| | The incidence will be calculated as number of patients with an AE, etc. or |
| | an ADR, etc./number of patients excluded from safety evaluation × 100. |
| | For PT, multiple episodes of the same ADR, etc. (PT) in the same patient will |
| | be tabulated as 1 patient/1 event to calculate the incidence as follows: |
| | [When safety is tabulated in patients included in safety evaluation] |
| | The incidence will be calculated as number of AE, etc. or ADR, |
| | etc./number of patients included in safety evaluation × 100. |
| | [When safety is tabulated in patients excluded from safety evaluation] |
| | The incidence will be calculated as number of AE, etc. or ADR, |
| | etc./number of patients excluded from safety evaluation × 100. |
| Time of onset | Time of onset will be calculated as date of onset of AE, etc. (or ADR, etc.) - |
| | start date of treatment + 1. |
| | If the month and day of AE, etc. (or ADR, etc.) is unknown, January 1 will be |
| | used for calculation. If an AE, etc. (or ADR, etc.) occurs in the same year as |
| | treatment is started, the month and day of starting treatment will be used for |
| | calculation. |
| | If the day of AE, etc. (or ADR, etc.) is unknown, 1 will be used for |
| | calculation. If an AE, etc. (or ADR, etc.) occurs in the same year and month |
| | as treatment is started, the start date of treatment will be used for calculation. |
| Patient with concurrent | Patient with a check for diabetes in the column of concurrent illness in the |
| diabetes | CRF or concurrent illness corresponding to SMQ code 20000041 |
| | (hyperglycaemia/new onset diabetes mellitus SMQ [scope: narrow]) |
| | described |
| Patient with concurrent | Patient with a check for dyslipidemia in the column of concurrent illness in |
| dyslipidemia | the CRF or concurrent illness corresponding to SMQ code 20000026 |
| | (dyslipidaemia SMQ [scope: narrow]) described |
| Patient with concurrent | Patient with a check for hyperuricemia in the column of concurrent illness in |
| hyperuricemia | the CRF or concurrent illness corresponding to MedDRA PT code 10020903 |

| Term | Definition |
|---|---|
| | (hyperuricaemia) described |
| Patient with concurrent coronary artery disease | Patient with a check for myocardial infarction or angina in the column of concurrent illness in the CRF, concurrent illness corresponding to SMQ code 20000043 (ischaemic heart disease SMQ [scope: narrow]) described in the column of other disease: name of disease, or PT corresponding to SMQ code 20000047 (myocardial infarction SMQ [scope: narrow]) described in the |
| Patient with concurrent | column of medical history Patient with a check for cardiac failure in the column of concurrent illness in |
| cardiac failure | the CRF or concurrent illness corresponding to SMQ code 20000004 (cardiac failure SMQ [scope: narrow]) described in the column of other disease: name of disease |
| Patient with concurrent myocardial infarction (including old myocardial infarction) | Patient with a check for myocardial infarction in the column of concurrent illness in the CRF or PT corresponding to SMQ code 20000047 (myocardial infarction SMQ [scope: narrow]) described in the column of other disease: name of disease or medical history |
| Patient with concurrent angina | Patient with a check for angina in the column of concurrent illness in the CRF or concurrent illness corresponding to MedDRA PT code 10002383 (angina pectoris), 10002388 (angina unstable), 10036759 (Prinzmetal angina), or 10058144 (postinfarction angina) described in the column of other disease: name of disease |
| Patient with concurrent coronary artery disease (other) | Patient with concurrent coronary artery disease who is not a patient with concurrent myocardial infarction (including old myocardial infarction) or angina |
| Patient with concurrent atrial fibrillation | Patient with a check for atrial fibrillation in the column of concurrent illness in the CRF or concurrent illness corresponding to MedDRA PT code 10003658 (atrial fibrillation) described in the column of other disease: name of disease |
| Patient with concurrent renal impairment | Patient with a check for chronic kidney disease (CKD), diabetic nephropathy, nephrosclerosis, or other in the column of concurrent illness in the CRF or concurrent illness corresponding to the following (1), (2), or (3) described in the column of other disease: name of disease: (1) SMQ code 20000213 (chronic kidney disease SMQ [scope: narrow]) (2) Takeda MedDRA query (hereinafter referred to as TMQ) (Renal Disease) (3) TMQ (Renal Impairment) |
| Patient with concurrent | Patient with a check for chronic kidney disease (CKD), diabetic nephropathy, |

| Term | Definition |
|---|---|
| chronic kidney disease | nephrosclerosis, or other in the column of concurrent illness in the CRF or |
| (CKD) | concurrent illness corresponding to SMQ code 20000213 (chronic kidney |
| | disease SMQ [scope: narrow]) described in the column of other disease: name |
| | of disease |
| Patient with concurrent | Patient with a check for diabetic nephropathy in the column of concurrent |
| diabetic nephropathy | illness in the CRF or concurrent illness corresponding to MedDRA PT code |
| | 10061835 (diabetic nephropathy) described in the column of other disease: |
| | name of disease |
| Patient with concurrent | Patient with a check for nephrosclerosis in the column of concurrent illness in |
| nephrosclerosis | the CRF or concurrent illness corresponding to MedDRA PT code 10029159 |
| | (nephrosclerosis) described in the column of other disease: name of disease |
| Patient with concurrent | Patient with concurrent chronic kidney disease (CKD) who is not a patient |
| chronic kidney disease | with concurrent diabetic nephropathy or nephrosclerosis |
| (CKD) (other) | |
| Patient with concurrent renal | Patient with concurrent renal impairment who is not a patient with concurrent |
| impairment (other) | chronic kidney disease (CKD), diabetic nephropathy, nephrosclerosis, or |
| | chronic kidney disease (CKD) (other) |
| Patient with concurrent | Patient with a check for hepatic steatosis or alcoholic hepatopathy in the |
| hepatic impairment | column of concurrent illness in the CRF or concurrent illness corresponding |
| | to the following (1), (2), or (3) described in the column of other disease: name |
| | of disease: |
| | (1) Standardised MedDRA query (hereinafter referred to as SMQ) code |
| | 20000005 (hepatic disorders SMQ [scope: narrow]) |
| | (2) MedDRA PT code 10019708 (hepatic steatosis) |
| | (3) MedDRA PT code 10001627 (alcoholic liver disease) |
| Patient with concurrent | Patient with a check for hepatic steatosis in the column of concurrent illness |
| hepatic steatosis | in the CRF or concurrent illness corresponding to MedDRA PT code |
| | 10019708 (hepatic steatosis) described in the column of other disease: name |
| | of disease |
| Patient with concurrent | Patient with a check for alcoholic hepatopathy in the column of concurrent |
| alcoholic hepatopathy | illness in the CRF or concurrent illness corresponding to MedDRA PT code |
| | 10001627 (alcoholic liver disease) described in the column of other disease: |
| | name of disease |
| Patient with concurrent | Patient with concurrent hepatic impairment who is not a patient with |
| hepatic impairment (other) | concurrent hepatic steatosis or alcoholic hepatopathy |
| Patient with concurrent | Patient with PT corresponding to SMQ code 20000060 (cerebrovascular |

| Term | Definition |
|---|---|
| cerebrovascular disorder | disorders SMQ [scope: narrow]) described in the column of concurrent |
| | illness: other disease: name of disease or medical history in the CRF |
| Age | If the month and day of starting treatment is smaller than the month and day |
| | of birth, age will be calculated as year of starting treatment - year of birth - 1. |
| | If the month and day of starting treatment is equal to or greater than the |
| | month and day of birth, age will be calculated as year of starting treatment - |
| | year of birth. |
| | If the month and day of birth is unknown, January 1 will be used for |
| | calculation. If the day of birth is unknown, 1 will be used for calculation. |
| Young, middle-aged, or | Patient aged 15 years or older and 74 years or younger |
| young-old patient | |
| Old-old patient | Patient aged 75 years or older |
| BMI | BMI will be calculated as body weight (kg) / [0.0001 × height (cm) × height |
| | (cm)]. BMI will be displayed to one decimal place by rounding. |
| Concomitant drug | Drug used during treatment with Zacras |
| Concomitant drug (at the | Concomitant drug that is started before the start of treatment with Zacras and |
| start of treatment with | is not terminated at the start of treatment with Zacras, or concomitant drug |
| Zacras) | that is started on the start day of treatment with Zacras |
| Concomitant drug (during | Concomitant drug used during a period from the start day of treatment with |
| the survey period) | Zacras to the end day of treatment with Zacras, including drugs used during |
| | the off-treatment period |
| Concomitant drug (at the end | Concomitant drug used on the end day of treatment with Zacras |
| of treatment with Zacras) | |
| Antihypertensive used | Drug described in the column for details on the use of other antihypertensive |
| within 2 months before the | in the CRF that is started before the start day of treatment with Zacras and |
| start of treatment with | used within 2 months (60 days) before the start of treatment with Zacras |
| Zacras | (excluding drugs that are started on the start day of treatment with Zacras) |
| Antidiabetic | Drugs with a NHI drug code starting with 396, 2492, or 249941 |
| Antidyslipidemic | Drugs with a NHI drug code starting with 218 or any of the following 7-digit |
| | numbers: |
| | 2190101, 2190102, 2190103, 2190104 |
| Antihyperuricemic | Drugs with a NHI drug code starting with 394 |
| Antihypertensive | ACE inhibitors, angiotensin receptor blockers (ARBs), diuretics (thiazide and |
| | thiazide analogue diuretics), calcium antagonists (Ca antagonists), direct |
| | renin inhibitors, aldosterone antagonists/potassium-sparing diuretics, |
| | vasodilators, β-blockers, central sympathetic inhibitors, αβ-blockers, |

| Term | Definition |
|---|---|
| | $\alpha_1$ -blockers, fixed-dose combination: ARB + diuretic, fixed-dose |
| | combination: ARB + calcium antagonist (Ca antagonist), and fixed-dose |
| | combination: calcium antagonist + statin in a list of antihypertensives in the |
| | Guidelines for the Management of Hypertension 2014 (JSH2014) |
| ACE inhibitor | Drugs described in the column for details on the use of other antihypertensive |
| | in the CRF that have a NHI drug code starting with the following 4-digit |
| | number: |
| | 2144 |
| | Generic name: captopril, enalapril maleate, perindopril erbumine, lisinopril |
| | hydrate, alacepril, delapril hydrochloride, benazepril hydrochloride, cilazapril |
| | hydrate, imidapril hydrochloride, temocapril hydrochloride, quinapril |
| | hydrochloride, trandolapril |
| ARB | Drugs described in the column for details on the use of other antihypertensive |
| | in the CRF that have a NHI drug code starting with any of the following |
| | 7-digit numbers: |
| | 2149039, 2149040, 2149041, 2149042, 2149044, 2149046, 2149048, |
| | 2149110, 2149111, 2149112, 2149113, 2149119, 2149116, 2149114, |
| | 2149117, 2149118, 2149115, 2149120, 2149121 |
| | Generic name: losartan potassium, candesartan cilexetil, valsartan, |
| | telmisartan, olmesartan medoxomil, irbesartan, azilsartan |
| Diuretic (thiazide and | Drugs described in the column for details on the use of other antihypertensive |
| thiazide analogue diuretic) | in the CRF that have a NHI drug code starting with any of the following |
| | 7-digit numbers: |
| | 2132003, 2132004, 2132006, 2149103, 2149012, 2135001, 2149007, |
| | 2149003, 2149110, 2149111, 2149112, 2149113, 2149119 |
| | Generic name: trichlormethiazide, hydrochlorothiazide, |
| | benzylhydrochlorothiazide, indapamide, mefruside, tripamide, meticrane, |
| | valsartan/hydrochlorothiazide, telmisartan/hydrochlorothiazide |
| HCTZ | Drugs described in the column for details on the use of other antihypertensive |
| | in the CRF that have a NHI drug code starting with any of the following |
| | 7-digit numbers: |
| | 2132004, 2149110, 2149111, 2149112, 2149113 |
| | Generic name: hydrochlorothiazide, losartan potassium/hydrochlorothiazide, |
| | candesartan cilexetil/hydrochlorothiazide, |
| Dose of HCTZ | The dose of HCTZ is the maximum dose in patients receiving HCTZ. |
| Ca antagonist | Drugs described in the column for details on the use of other antihypertensive |

| Term | Definition |
|---|---|
| | in the CRF that have a NHI drug code starting with any of the following |
| | 7-digit numbers: |
| | 2171022, 2171014, 2171019, 2171020, 2149019, 2149022, 2149043, |
| | 2149027, 2149034, 2149037, 2149038, 2171021, 2149035, 2149030, |
| | 2171006, 2149116, 2149114, 2149117, 2149118, 2149115, 2190101, |
| | 2190102, 2190103, 2190104, 2149120, 2149121 |
| | Generic name: amlodipine besilate, nifedipine, nisoldipine, nitrendipine, |
| | nicardipine hydrochloride, nilvadipine, azelnidipine, manidipine |
| | hydrochloride, efonidipine hydrochloride ethanol, cilnidipine, aranidipine, |
| | benidipine hydrochloride, felodipine, barnidipine hydrochloride, diltiazem |
| | hydrochloride |
| Direct renin inhibitor | Drugs described in the column for details on the use of other antihypertensive |
| | in the CRF that have a NHI drug code starting with the following 7-digit |
| | number: |
| | 2149047 |
| | Generic name: aliskiren fumarate |
| Aldosterone | Drugs described in the column for details on the use of other antihypertensive |
| antagonist/potassium-sparing | in the CRF that have a NHI drug code starting with any of the following |
| diuretic | 7-digit numbers: |
| | 2133001, 2149045, 2133002 |
| | Generic name: spironolactone, eplerenone, triamterene |
| Aldosterone antagonist | Drugs described in the column for details on the use of other antihypertensive |
| | in the CRF that have a NHI drug code starting with any of the following |
| | 7-digit numbers: |
| | 2133001, 2149045, |
| | Generic name: spironolactone, eplerenone |
| Potassium-sparing diuretic | Drugs described in the column for details on the use of other antihypertensive |
| | in the CRF that have a NHI drug code starting with the following 7-digit |
| | number: |
| | 2133002 |
| | Generic name: triamterene |
| Diuretic | Diuretics (thiazide and thiazide analogue diuretics) or potassium-sparing |
| | diuretics described in the column for details on the use of other |
| | antihypertensive in the CRF |
| Vasodilator | Drugs described in the column for details on the use of other antihypertensive |
| | in the CRF that have a NHI drug code starting with the following 7-digit |

| Term | Definition |
|---|---|
| | number: |
| | 2142004 |
| | Generic name: hydralazine hydrochloride |
| β-blocker | Drugs described in the column for details on the use of other antihypertensive |
| | in the CRF that have a NHI drug code starting with any of the following |
| | 7-digit numbers: |
| | 2123011, 2123016, 2149700, 2149031, 2149010, 2123001, 2149029, |
| | 2123008, 2149014, 2149021, 2149028, 2123015, 2123005, 2149025, |
| | 2123009, 2149011 |
| | Generic name: atenolol, bisoprolol fumarate, bisoprolol, betaxolol |
| | hydrochloride, metoprolol tartrate, acebutolol hydrochloride, celiprolol |
| | hydrochloride, propranolol hydrochloride, nipradilol, tilisolol hydrochloride, |
| | nadolol, carteolol hydrochloride, pindolol |
| Central sympathetic inhibitor | Drugs described in the column for details on the use of other antihypertensive |
| | in the CRF that have a NHI drug code starting with any of the following |
| | 7-digit numbers: |
| | 2149001, 2149017, 2145001 |
| | Generic name: clonidine hydrochloride, guanabenz acetate, methyldopa |
| | hydrate |
| αβ-blocker | Drugs described in the column for details on the use of other antihypertensive |
| | in the CRF that have a NHI drug code starting with any of the following |
| | 7-digit numbers: |
| | 2149032, 2149018, 2123014, 2149009, 2149036 |
| | Generic name: carvedilol, amosulalol hydrochloride, arotinolol |
| | hydrochloride, labetalol hydrochloride, bevantolol hydrochloride |
| $\alpha_1$ -blocker | Drugs described in the column for details on the use of other antihypertensive |
| | in the CRF that have a NHI drug code starting with any of the following |
| | 7-digit numbers: |
| | 2149026, 2149015, 2149023, 2149002, 2149020 |
| | Generic name: doxazosin mesilate, bunazosin hydrochloride, terazosin |
| | hydrochloride hydrate, prazosin hydrochloride, urapidil |
| Fixed-dose combination: | Drugs described in the column for details on the use of other antihypertensive |
| ARB + diuretic | in the CRF that have a NHI drug code starting with any of the following |
| | 7-digit numbers: |
| | 2149110, 2149111, 2149112, 2149113, 2149119 |
| | Generic name: losartan potassium/hydrochlorothiazide, candesartan |

| Term | Definition |
|---|---|
| | cilexetil/hydrochlorothiazide, valsartan/hydrochlorothiazide, |
| | telmisartan/hydrochlorothiazide, irbesartan/trichlormethiazide |
| Fixed-dose combination: | Drugs described in the column for details on the use of other antihypertensive |
| ARB + Ca antagonist | in the CRF that have a NHI drug code starting with any of the following |
| | 7-digit numbers: |
| | 2149116, 2149114, 2149117, 2149118, 2149115, 2149120 |
| | Generic name: candesartan cilexetil/amlodipine besilate, valsartan/amlodipine |
| | besilate, telmisartan/amlodipine besilate, irbesartan/amlodipine besilate, |
| | olmesartan medoxomil/azelnidipine, valsartan/cilnidipine |
| Fixed-dose combination: Ca | Drugs described in the column for details on the use of other antihypertensive |
| antagonist + statin | in the CRF that have a NHI drug code starting with any of the following |
| | 7-digit numbers: |
| | 2190101, 2190102, 2190103, 2190104 |
| | Generic name: amlodipine besilate/atorvastatin calcium hydrate |
| Other (antihypertensive) | Vasodilators, β-blockers, central sympathetic inhibitors, αβ-blockers, and |
| | $\alpha_1$ -blockers described in the column for details on the use of other |
| | antihypertensive in the CRF |
| Number of concomitant | The number of drugs described in the column for details on the use of other |
| drugs (antihypertensive other | antihypertensive in the CRF will be tabulated. The fixed-dose combination |
| than Zacras) | will be tabulated as one drug. For instance, "fixed-dose combination: ARB + |
| | diuretic" used concomitantly will be tabulated as one drug. |
| eGFR (mL/min/1.73 m <sup>2</sup> ) | eGFR will be calculated as 194 × serum creatinine [mg/dL] <sup>-1.094</sup> × age |
| | [years] <sup>-0.287</sup> (× 0.739 for females). eGFR will be displayed as an integer by |
| | rounding. |
| Summary statistics | Mean, standard deviation, minimum, first quartile, median, third quartile, |
| | maximum |

# 1.2 Number of Digits to be Displayed

| Term | Definition |
|--------------------|--------------------------------------------------------|
| Percentage (%) | Incidence of AE, etc. or ADR, etc.: |
| | Displayed to two decimal places by rounding |
| | Other: |
| | Displayed to one decimal place by rounding |
| Summary statistics | Mean: |
| (mean/standard | Displayed to one lower digit than raw data by rounding |
| deviation) | Standard deviation: |

| Term | Definition |
|---|---|
| | Displayed to two lower digits than raw data by rounding |
| P-value | P-value will be displayed to three decimal places by rounding down. |
| | P-value rounded down to less than 0.001 will be displayed as p<0.001. |

#### 1.3 Level of Significance

Two-sided 5%

#### 1.4 Handling of Test/Measurement Data

Test/measurement data will be handled in accordance with the criteria described below (with 1 month as 30 days). If there are multiple pieces of data at the same specified time point, data on the test day closest to the specified day of assessment will be employed, and the latest data among different pieces of data on different days with the same deviation from the specified day of assessment will be employed. At the final assessment\*, values measured on the day closest to the start date of treatment with Zacras + 375 days will be employed (including values measured during the off-treatment period). Values measured after the end day of treatment with Zacras will not be employed.

The number of days from the start day of treatment with Zacras is 1 day for the start day of treatment with Zacras and -1 day for the previous day.

\* After 12 months of treatment with Zacras (or at discontinuation of treatment with Zacras)

| Time point of test | Permissible range (number of days from the start day of treatment) | Specified day of assessment |
|---|---|---|
| At the start of treatment | -90 to -1 | Start date of treatment |
| After 1 month of treatment | 1 to 45 | Start date of treatment + 30 |
| After 2 months of treatment | 46 to 75 | Start date of treatment + 60 |
| After 3 months of treatment | 76 to 105 | Start date of treatment + 90 |
| After 4 months of treatment | 106 to 135 | Start date of treatment + 120 |
| After 5 months of treatment | 136 to 165 | Start date of treatment + 150 |
| After 6 months of treatment | 166 to 195 | Start date of treatment + 180 |
| After 7 months of treatment | 196 to 225 | Start date of treatment + 210 |
| After 8 months of treatment | 226 to 255 | Start date of treatment + 240 |
| After 9 months of treatment | 256 to 285 | Start date of treatment + 270 |
| After 10 months of treatment | 286 to 315 | Start date of treatment + 300 |
| After 11 months of treatment | 316 to 345 | Start date of treatment + 330 |
| After 12 months of treatment | 346 to 375 | Start date of treatment + 360 |

| At the final assessment | 1 to 375 | Start date of treatment + |
|-------------------------|----------|---------------------------|
| | | 3/5 |

#### 2.0 Disposition of Patients (Patient Composition Diagram)

(1) Patients included in tabulation/analysis

Patients enrolled in the specified drug-use survey

#### (2) Data tabulated/analyzed

The number of enrolled patients, number of medical institutions involved in patient registration, number of patients from whom the CRF is collected, number of patients from whom the CRF is not collected, number of finalized patients, number of non-finalized patients, number of patients included in safety evaluation, number of patients excluded from safety evaluation, number of patients included in efficacy evaluation, and number of patients excluded from efficacy evaluation will be tabulated.

For the number of medical institutions involved in patient registration, one medical institution with different departments should not be counted more than once.

For patients from whom the CRF is not collected, the number of patients by reason for failure to collect and the total number will be tabulated.

For patients excluded from safety evaluation and those excluded from efficacy evaluation, the number of patients by reason for exclusion and the total number will be tabulated.

Patients meeting any of the criteria listed below will be handled as described below regarding whether to employ them or not.

| Criterion | Enrollment | Safety<br>evaluation | Efficacy evaluation |
|---|---|---|---|
| Duplicate registration (the same patient) | × | - | - |
| [posterior finding] | | | |
| Wrong registration (not prescribed) [posterior | × | - | - |
| finding] | | | |
| Treatment before the contract period [posterior | 0 | × | × |
| finding] | | | |
| Registration after 15 days of treatment with | 0 | × | × |
| Zacras [posterior finding] | | | |
| No data on blood pressure before or after | 0 | 0 | × |
| treatment with Zacras | | | |
| Deviation from inclusion criteria | 0 | 0 | × |
| Deviation from exclusion criteria | 0 | 0 | × |
| Failure to confirm the intake of Zacras [during | × | - | - |
| the patient enrollment period] | | | |
| Failure to confirm the intake of Zacras [after | 0 | × | × |
| the patient enrollment period] | | | |

| Unavailability of follow-up CRF | 0 | 0 | 0 |
|---------------------------------|---|---|---|
|---------------------------------|---|---|---|

o: employed, ×: excluded or not employed

# (3) Table/figure number

Figure 2.0-1, Table 2.0-1

# 3.0 Patient Demographics and Baseline Characteristics

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

## (2) Data tabulated/analyzed

For each variable, patients will be categorized as described below, and the number and proportion of patients will be tabulated.

| Variable | Category |
|---|---|
| Sex | Male, female |
| Age | Summary statistics |
| | <65 years, ≥65 years |
| | <65 years, 65 to 74 years, ≥75 years |
| Duration of disease | <1 year, 1 to <3 years, 3 to <5 years, ≥5 years, unknown |
| Diagnostic category | |
| (at the start of | Outpatient, inpatient |
| treatment with Zacras) | |
| Predisposition to | No, yes, unknown |
| hypersensitivity | 10, yes, anknown |
| Concurrent illness | No, yes |
| | Diabetes, dyslipidemia, hyperuricemia, cardiac failure, coronary artery |
| Disposition | disease (myocardial infarction (including old myocardial infarction), |
| (multiple | angina, or other), atrial fibrillation, renal impairment (chronic kidney |
| tabulation) | disease (CKD) [diabetic nephropathy, nephrosclerosis, or other] or |
| | other), hepatic impairment (hepatic steatosis, alcoholic hepatopathy, or |
| | other), cerebrovascular disorder |
| Medical history | No, yes, unknown |
| Body weight (kg) | Summary statistics |
| | $<40, 40 \text{ to } <50, 50 \text{ to } <60, 60 \text{ to } <70, \ge 70, \text{ not measured}$ |
| BMI (kg/m <sup>2</sup> ) | Summary statistics |
| | <18.5, 18.5 to <25.0, 25.0 to <30.0, ≥30.0, unknown |
| eGFR [at the start of | Summary statistics |
| treatment] | <15, 15 to <30, 30 to <45, 45 to <60, 60 to <90, ≥90, unknown |
| (mL/min/1.73 m <sup>2</sup> ) | 10, 10 to 20, 20 to 10, 10 to 00, 00 to 30, _30, _amazona |
| Smoking history | Never smoked, current smoker, past smoker, unknown |
| Drinking history | |
| (drink alcoholic | Yes, no, unknown |
| beverage almost every | |
| day) | |

| Presence or absence | |
|------------------------|---------|
| of breast-feeding (at | |
| the start of treatment | No, yes |
| with Zacras) [only | |
| females] | |

Table 3.0-1

## 4.0 Treatment Given

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

## (2) Data tabulated/analyzed

For each variable, patients will be categorized as described below, and the number and proportion of patients will be tabulated.

| Variable | Category |
|---|---|
| Initial dose of Zacras | LD, HD |
| Presence or absence | |
| of change in daily | No, yes |
| dose of Zacras | |
| Disposition | $LD \rightarrow HD, HD \rightarrow LD$ |
| Duration of treatment | 1 to 190 days 191 to 260 days >261 days |
| with Zacras | 1 to 180 days, 181 to 360 days, ≥361 days |
| Presence or absence | |
| of discontinuation of | No, yes |
| treatment with Zacras | |
| Reason for | Successful achievement of treatment goal, AE, patient's failure to visit |
| discontinuation of | the hospital such as transfer to another hospital, insufficient efficacy, |
| treatment with Zacras | other |
| Treatment with | |
| antihypertensive other | |
| than Zacras (at the | No, yes |
| start of treatment with | |
| Zacras) | |
| | ACE inhibitor, ARB, diuretic (thiazide and thiazide analogue diuretic), |
| Disposition (multiple | Ca antagonist, direct renin inhibitor, aldosterone antagonist, |
| tabulation)* | potassium-sparing diuretic, fixed-dose combination: ARB + diuretic, |
| | fixed-dose combination: ARB + Ca antagonist, fixed-dose combination: |
| | calcium antagonist + statin, other |
| Antihypertensive | |
| other than Zacras: | |
| treatment with HCTZ | No, yes |
| (at the start of | |
| treatment with Zacras) | |
| Disposition | 6.25 mg, 12.5 mg, other |
| Treatment with | No, yes |

| antihypertensive other<br>than Zacras (during<br>the survey period) | |
|---|---|
| Disposition (multiple tabulation)* | ACE inhibitor, ARB, diuretic (thiazide and thiazide analogue diuretic), Ca antagonist, direct renin inhibitor, aldosterone antagonist, potassium-sparing diuretic, fixed-dose combination: ARB + diuretic, fixed-dose combination: ARB + Ca antagonist, fixed-dose combination: calcium antagonist + statin, other |
| Antihypertensive other than Zacras: treatment with HCTZ (during the survey period) | No, yes |
| Disposition | 6.25 mg, 12.5 mg, other |
| Treatment with antihypertensive other than Zacras (within 2 months before the start of treatment with Zacras) | No, yes |
| Disposition (multiple tabulation)* | ACE inhibitor, ARB, diuretic (thiazide and thiazide analogue diuretic), Ca antagonist, direct renin inhibitor, aldosterone antagonist, potassium-sparing diuretic, fixed-dose combination: ARB + diuretic, fixed-dose combination: ARB + Ca antagonist, fixed-dose combination: calcium antagonist + statin, other |
| Number of concomitant drugs (antihypertensive other than Zacras) | |
| (at the start of treatment with Zacras) | 0, 1, 2, 3, 4, 5, ≥6 |
| (at the end of treatment with Zacras) | 0, 1, 2, 3, 4, 5, ≥6 |
| Concomitant non-antihypertensive drug (during the survey period) | No, yes |

| Disposition | |
|-------------|----------------------------------------------------------|
| (multiple | Antidiabetic, antidyslipidemic, antihyperuricemic, other |
| tabulation) | |

<sup>\*</sup> For fixed-dose combinations, individual ingredients will be tabulated separately. If "fixed-dose combination: ARB + diuretic" is used concomitantly, for instance, "ARB" and "diuretic" will also be tabulated.

Table 4.0-1

#### 5.0 Tabulation/Analysis of Safety

#### 5.1 Occurrence of Adverse Events/Infections and Adverse Drug Reactions/Infections

#### 5.1.1 Occurrence of Adverse Events/Infections

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with | N. I. C. C. A. I. A. F. A. |
| an AE, etc. | Number of patients who experienced an AE, etc. |
| | Number of reported AE, etc. Multiple episodes of the same AE, etc. |
| Number of AE, etc. | (PT) in the same patient will be tabulated as the total number of |
| | episodes. |
| | The incidence of AE, etc. will be calculated as number of patients |
| Incidence of AE, etc. | with an AE, etc./number of patients included in safety evaluation $\times$ |
| | 100. |
| | AEs, etc. will be classified by SOC and then tabulated by PT. For |
| | laboratory tests, AEs, etc. will be classified by SOC, then sorted by |
| | HLGT, and finally tabulated by PT. |
| Tyme of A.E. ata | For SOC, the number of patients with an AE, etc. and the incidence |
| Type of AE, etc. | of AE, etc. will be listed by SOC internationally agreed order. |
| | For PT, the number and incidence of AE, etc. will be listed in |
| | ascending order of PT code. Multiple episodes of the same AE, etc. |
| | (PT) in the same patient will be tabulated as 1 patient/1 event. |

#### (3) Table/figure number

Table 5.1-1

#### 5.1.2 Occurrence of Adverse Drug Reactions/Infections

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with an ADR, etc. | Number of patients who experienced an ADR, etc. |
| Number of ADR, etc. | Number of reported ADR, etc. Multiple episodes of the same ADR, etc. (PT) in the same patient will be tabulated as the total number of |

| | episodes. |
|---|---|
| Incidence of ADR, etc. | The incidence of ADR, etc. will be calculated as number of patients |
| | with an ADR, etc./number of patients included in safety evaluation |
| | × 100. |
| | ADRs, etc. will be classified by SOC and then tabulated by PT. For |
| | laboratory tests, ADRs, etc. will be classified by SOC, then sorted |
| | by HLGT, and finally tabulated by PT. |
| | For SOC, the number of patients with an ADR, etc. and the |
| Type of ADR, etc. | incidence of ADR, etc. will be listed by SOC internationally agreed |
| | order. |
| | For PT, the number and incidence of ADR, etc. will be listed in |
| | ascending order of PT code. Multiple episodes of the same ADR, |
| | etc. (PT) in the same patient will be tabulated as 1 patient/1 event. |

Table 5.1-2

- 5.2 Occurrence of Adverse Events/Infections and Adverse Drug Reactions/Infections in Patients Excluded from Safety Evaluation
  - 5.2.1 Occurrence of Adverse Events/Infections
    - (1) Patients included in tabulation/analysis

      Patients excluded from safety evaluation
    - (2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with | Number of patients who experienced an AE, etc. |
| an AE, etc. | 1 / |
| | Number of reported AE, etc. Multiple episodes of the same AE, etc. |
| Number of AE, etc. | (PT) in the same patient will be tabulated as the total number of |
| | episodes. |
| Incidence of AE, etc. | The incidence of AE, etc. will be calculated as number of patients |
| | with an AE, etc./number of patients excluded from safety evaluation |
| | × 100. |
| Type of AE, etc. | AEs, etc. will be classified by SOC and then tabulated by PT. For |
| | laboratory tests, AEs, etc. will be classified by SOC, then sorted by |
| | HLGT, and finally tabulated by PT. |
| | For SOC, the number of patients with an AE, etc. and the incidence |
| | of AE, etc. will be listed by SOC internationally agreed order. |

| For PT, the number and incidence of AE, etc. will be listed in |
|--------------------------------------------------------------------|
| ascending order of PT code. Multiple episodes of the same AE, etc. |
| (PT) in the same patient will be tabulated as 1 patient/1 event. |

Table 5.2-1

#### 5.2.2 Occurrence of Adverse Drug Reactions/Infections

(1) Patients included in tabulation/analysis

Patients excluded from safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with an ADR, etc. | Number of patients who experienced an ADR, etc. |
| Number of ADR, etc. | Number of reported ADR, etc. Multiple episodes of the same ADR, etc. (PT) in the same patient will be tabulated as the total number of episodes. |
| Incidence of ADR, etc. | The incidence of ADR, etc. will be calculated as number of patients with an ADR, etc./number of patients excluded from safety evaluation × 100. |
| Type of ADR, etc. | ADRs, etc. will be classified by SOC and then tabulated by PT. For laboratory tests, ADRs, etc. will be classified by SOC, then sorted by HLGT, and finally tabulated by PT. For SOC, the number of patients with an ADR, etc. and the incidence of ADR, etc. will be listed by SOC internationally agreed order. For PT, the number and incidence of ADR, etc. will be listed in ascending order of PT code. Multiple episodes of the same ADR, etc. (PT) in the same patient will be tabulated as 1 patient/1 event. |

(3) Table/figure number

Table 5.2-2

- 5.3 Occurrence of Adverse Events/Infections and Adverse Drug Reactions/Infections by Seriousness, Time of Onset, and Outcome
  - 5.3.1 Occurrence of Adverse Events/Infections by Seriousness, Time of Onset, and Outcome
    - (1) Patients included in tabulation/analysis

Patients included in safety evaluation

#### (2) Data tabulated/analyzed

AEs, etc. will be categorized for each variable as described below, and the type of AE, etc. will be tabulated.

| Variable | Category |
|---|---|
| Seriousness | Serious, non-serious |
| Time of onset | Days 1 to 180, Days 181 to 360, Day 361 or later |
| Outcome | Recovered, recovering, not recovered, recovered with sequelae, fatal, unknown |

The type of AE, etc. will be tabulated as described below.

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients | Number of patients who experienced an AE, etc. by SOC/PT |
| Number of AE, etc. | Number of reported AE, etc. by SOC/PT |
| | AEs, etc. will be classified by SOC and then tabulated by PT. For |
| | laboratory tests, AEs, etc. will be classified by SOC, then sorted by |
| | HLGT, and finally tabulated by PT. |
| | AEs, etc. will be listed for SOC by SOC internationally agreed |
| True of AE ato | order and for PT in ascending order of PT code. |
| Type of AE, etc. | Multiple episodes of the same AE, etc. (PT) in the same patient will |
| | be tabulated by category as the total number of episodes (for |
| | instance, one episode of serious diarrhoea and one episode of |
| | non-serious diarrhoea in the same patient will be counted once in |
| | the respective categories). |

#### (3) Table/figure number

Table 5.3-1

# 5.3.2 Occurrence of Adverse Drug Reactions/Infections by Seriousness, Time of Onset, and Outcome

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

ADRs, etc. will be categorized for each variable as described below, and the type of ADR, etc. will be tabulated.

| Variable | Category |
|---|---|
| Seriousness | Serious, non-serious |
| Time of onset | Days 1 to 180, Days 181 to 360, Day 361 or later |
| Outcome | Recovered, recovering, not recovered, recovered with sequelae, fatal, unknown |

The type of ADR, etc. will be tabulated as described below.

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients | Number of patients who experienced an ADR, etc. by SOC/PT |
| Number of ADR, etc. | Number of reported ADR, etc. by SOC/PT |
| | ADRs, etc. will be classified by SOC and then tabulated by PT. For |
| | laboratory tests, ADRs, etc. will be classified by SOC, then sorted |
| | by HLGT, and finally tabulated by PT. |
| | ADRs, etc. will be listed for SOC by SOC internationally agreed |
| Tyme of ADD ata | order and for PT in ascending order of PT code. |
| Type of ADR, etc. | Multiple episodes of the same ADR, etc. (PT) in the same patient |
| | will be tabulated by category as the total number of episodes (for |
| | instance, one episode of serious diarrhoea and one episode of |
| | non-serious diarrhoea in the same patient will be counted once in |
| | the respective categories). |

Table 5.3-2

- 5.4 Incidence of Adverse Event/Infection and Adverse Drug Reaction/Infection by Factors Related to Patient Demographics and Baseline Characteristics and Treatment Given
- 5.4.1 Incidence of Adverse Event/Infection by Factors Related to Patient Demographics and Baseline Characteristics and Treatment Given
  - (1) Patients included in tabulation/analysis

    Patients included in safety evaluation
  - (2) Data tabulated/analyzed

AEs, etc. will be categorized for each variable as described below, and the incidence of AE, etc. (point estimate and 95% CI) will be tabulated.

In addition, Fisher's exact probability test will be performed for variables with unranked categories, and the Mann-Whitney U test will be performed for variables with ranked categories.

| Variable | Category |
|--------------------|--------------------------------------|
| Sex | Male, female |
| Aga | <65 years, ≥65 years |
| Age | <65 years, 65 to 74 years, ≥75 years |
| Predisposition to | No voc unknown |
| hypersensitivity | No, yes, unknown |
| Concurrent illness | No, yes |

| Disposition<br>(multiple<br>tabulation) | Diabetes, dyslipidemia, hyperuricemia, cardiac failure, coronary artery disease (myocardial infarction (including old myocardial infarction), angina, or other), atrial fibrillation, renal impairment (chronic kidney disease (CKD) [diabetic nephropathy, nephrosclerosis, or other] or other), hepatic impairment (hepatic steatosis, alcoholic hepatopathy, or other), cerebrovascular disorder |
|---|---|
| Medical history | No, yes, unknown |
| Body weight (kg) | <40, 40 to <50, 50 to <60, 60 to <70, ≥70, not measured |
| BMI (kg/m <sup>2</sup> ) | <18.5, 18.5 to <25.0, 25.0 to <30.0, ≥30.0, unknown |
| Initial dose of Zacras | LD, HD |
| Presence or absence of change in daily dose of Zacras | No, yes |
| Disposition | $LD \rightarrow HD, HD \rightarrow LD$ |
| Duration of treatment with Zacras | 1 to 180 days, 181 to 360 days, ≥361 days The denominator is the number of patients treated with Zacras for 1 day or more to calculate the incidence of AE, etc. for "1 to x days" and the number of patients treated with Zacras for x + 1 days or more to calculate the incidence of AE, etc. for "x + 1 to y days." |
| Treatment with antihypertensive other than Zacras (at the start of treatment with Zacras) | No, yes |
| Disposition (multiple tabulation)* | ACE inhibitor, ARB, diuretic (thiazide and thiazide analogue diuretic), Ca antagonist, direct renin inhibitor, aldosterone antagonist, potassium-sparing diuretic, fixed-dose combination: ARB + diuretic, fixed-dose combination: ARB + Ca antagonist, fixed-dose combination: calcium antagonist + statin, other |
| Treatment with antihypertensive other than Zacras (during the survey period) | No, yes |
| Disposition (multiple tabulation)* | ACE inhibitor, ARB, diuretic (thiazide and thiazide analogue diuretic), Ca antagonist, direct renin inhibitor, aldosterone antagonist, potassium-sparing diuretic, fixed-dose combination: ARB + diuretic, fixed-dose combination: |

| | calcium antagonist + statin, other |
|---|---|
| Treatment with antihypertensive other than Zacras (within 2 months before the start of treatment with Zacras) | No, yes |
| Disposition (multiple tabulation)* | ACE inhibitor, ARB, diuretic (thiazide and thiazide analogue diuretic), Ca antagonist, direct renin inhibitor, aldosterone antagonist, potassium-sparing diuretic, fixed-dose combination: ARB + diuretic, fixed-dose combination: ARB + Ca antagonist, fixed-dose combination: calcium antagonist + statin, other |
| Concomitant non-antihypertensive drug (during the survey period) | No, yes |
| Disposition (multiple tabulation) | Antidiabetic, antidyslipidemic, antihyperuricemic, other |

<sup>\*</sup> For fixed-dose combinations, individual ingredients will be tabulated separately. If "fixed-dose combination: ARB + diuretic" is used concomitantly, for instance, "ARB" and "diuretic" will also be tabulated.

Table 5.4-1

# 5.4.2 Incidence of Adverse Drug Reaction/Infection by Factors Related to Patient Demographics and Baseline Characteristics and Treatment Given

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

#### (2) Data tabulated/analyzed

ADRs, etc. will be categorized for each variable as described below, and the incidence of ADR, etc. (point estimate and 95% CI) will be tabulated.

In addition, Fisher's exact probability test will be performed for variables with unranked categories, and the Mann-Whitney U test will be performed for variables with ranked categories.

| Variable | Category |
|----------|----------|
|----------|----------|

| Sex | Male, female |
|---|---|
| Age | <65 years, ≥65 years |
| | <65 years, 65 to 74 years, ≥75 years |
| Predisposition to | No, yes, unknown |
| hypersensitivity | ivo, yes, unknown |
| Concurrent illness | No, yes |
| | Diabetes, dyslipidemia, hyperuricemia, cardiac failure, coronary artery |
| | disease (myocardial infarction (including old myocardial infarction), |
| Disposition | angina, or other), atrial fibrillation, renal impairment (chronic kidney |
| Disposition | disease (CKD) [diabetic nephropathy, nephrosclerosis, or other] or |
| | other), hepatic impairment (hepatic steatosis, alcoholic hepatopathy, or |
| | other), cerebrovascular disorder |
| Medical history | No, yes, unknown |
| Body weight (kg) | <40, 40 to <50, 50 to <60, 60 to <70, ≥70, not measured |
| BMI (kg/m <sup>2</sup> ) | <18.5, 18.5 to <25.0, 25.0 to <30.0, ≥30.0, unknown |
| Initial dose of Zacras | LD, HD |
| Presence or absence | |
| of change in daily | No, yes |
| dose of Zacras | |
| Disposition | $LD \rightarrow HD, HD \rightarrow LD$ |
| | 1 to 180 days, 181 to 360 days, ≥361 days |
| Duration of treatment with Zacras | The denominator is the number of patients treated with Zacras for 1 day |
| | or more to calculate the incidence of AE, etc. for "1 to x days" and the |
| | number of patients treated with Zacras for $x + 1$ days or more to |
| | calculate the incidence of AE, etc. for "x + 1 to y days." |
| Treatment with | |
| antihypertensive other | |
| than Zacras (at the | No, yes |
| start of treatment with | |
| Zacras) | |
| | ACE inhibitor, ARB, diuretic (thiazide and thiazide analogue diuretic), |
| Disposition (multiple tabulation)* | Ca antagonist, direct renin inhibitor, aldosterone antagonist, |
| | potassium-sparing diuretic, fixed-dose combination: ARB + diuretic, |
| | fixed-dose combination: ARB + Ca antagonist, fixed-dose combination: |
| | calcium antagonist + statin, other |
| Treatment with | No, yes |
| antihypertensive other | |

| than Zacras (during | |
|---|---|
| the survey period) | |
| Disposition (multiple tabulation)* | ACE inhibitor, ARB, diuretic (thiazide and thiazide analogue diuretic), Ca antagonist, direct renin inhibitor, aldosterone antagonist, potassium-sparing diuretic, fixed-dose combination: ARB + diuretic, fixed-dose combination: ARB + Ca antagonist, fixed-dose combination: calcium antagonist + statin, other |
| Treatment with antihypertensive other than Zacras (within 2 months before the start of treatment with Zacras) | No, yes |
| Disposition (multiple tabulation)* | ACE inhibitor, ARB, diuretic (thiazide and thiazide analogue diuretic), Ca antagonist, direct renin inhibitor, aldosterone antagonist, potassium-sparing diuretic, fixed-dose combination: ARB + diuretic, fixed-dose combination: ARB + Ca antagonist, fixed-dose combination: calcium antagonist + statin, other |
| Concomitant non-antihypertensive drug (during the survey period) | No, yes |
| Disposition (multiple tabulation) | Antidiabetic, antidyslipidemic, antihyperuricemic, other |

<sup>\*</sup> For fixed-dose combinations, individual ingredients will be tabulated separately. If "fixed-dose combination: ARB + diuretic" is used concomitantly, for instance, "ARB" and "diuretic" will also be tabulated.

Table 5.4-2

- 5.5 Occurrence of Adverse Events/Infections and Adverse Drug Reactions/Infections by Age Group
  - 5.5.1 Occurrence of Adverse Events/Infections by Age Group
    - (1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The type of AE, etc. will be tabulated by age group (<65 years, 65 to 74 years,  $\ge 75$  years).

The type of AE, etc. will be tabulated as described in Section 5.1.

(3) Table/figure number

Table 5.5-1

#### 5.5.2 Occurrence of Adverse Drug Reactions/Infections by Age Group

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The type of ADR, etc. will be tabulated by age group (<65 years, 65 to 74 years,  $\ge 75$  years).

The type of ADR, etc. will be tabulated as described in Section 5.1.

(3) Table/figure number

Table 5.5-2

- 5.6 Occurrence of Adverse Events/Infections and Adverse Drug Reactions/Infections by the Presence or Absence of Concurrent Hepatic Impairment
  - 5.6.1 Occurrence of Adverse Events/Infections by the Presence or Absence of Concurrent Hepatic Impairment
    - (1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The type of AE, etc. will be tabulated by the presence or absence of concurrent hepatic impairment.

The type of AE, etc. will be tabulated as described in Section 5.1.

(3) Table/figure number

Table 5.6-1

- 5.6.2 Occurrence of Adverse Drug Reactions/Infections by the Presence or Absence of Concurrent Hepatic Impairment
  - (1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The type of ADR, etc. will be tabulated by the presence or absence of concurrent hepatic impairment.

The type of ADR, etc. will be tabulated as described in Section 5.1.

(3) Table/figure number

Table 5.6-2

5.7 Occurrence of Adverse Events/Infections and Adverse Drug Reactions/Infections by the Presence or

Absence of Concurrent Renal Impairment

# 5.7.1 Occurrence of Adverse Events/Infections by the Presence or Absence of Concurrent Renal Impairment

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The type of AE, etc. will be tabulated by the presence or absence of concurrent renal impairment.

The type of AE, etc. will be tabulated as described in Section 5.1.

(3) Table/figure number

Table 5.7-1

# 5.7.2 Occurrence of Adverse Drug Reactions/Infections by the Presence or Absence of Concurrent Renal Impairment

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The type of ADR, etc. will be tabulated by the presence or absence of concurrent renal impairment.

The type of ADR, etc. will be tabulated as described in Section 5.1.

(3) Table/figure number

Table 5.7-2

- 5.8 Occurrence of Adverse Drug Reactions/Infections by the Presence or Absence of Concomitant Antihypertensive Other than Zacras (during the Survey Period)
  - (1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The type of ADR, etc. will be tabulated by the presence or absence of concomitant antihypertensive other than Zacras (during the survey period).

The type of ADR, etc. will be tabulated as described in Section 5.1.

A patient with "yes" for concomitant antihypertensive other than Zacras (during the survey period) and an ADR, etc. will be handled as a patient with "no" for concomitant antihypertensive other than Zacras if the ADR, etc. occurs before the start of concomitant treatment. A patient with "yes" for concomitant antihypertensive other than Zacras (during the survey period) and multiple ADRs, etc. will be handled as a patient with "yes" for concomitant antihypertensive other than Zacras if at least one ADR, etc. occurs after the start of concomitant treatment

(3) Table/figure number
Table 5.8

#### 5.9 Listing of Occurrence of Serious Adverse Events/Infections

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---|---|
| Number of patients with a | Number of patients who experienced a SAE, etc. |
| SAE, etc. | Number of patients who experienced a SAE, etc. |
| | Number of reported SAE, etc. |
| Number of SAE, etc. | Multiple episodes of the same SAE, etc. (PT) in the same patient |
| | will be tabulated as the total number of episodes. |
| | The incidence of SAE, etc. will be calculated as number of patients |
| Incidence of SAE, etc. | with a SAE, etc./number of patients included in safety evaluation × |
| | 100. |
| | SAEs, etc. will be classified by SOC and then tabulated by PT. For |
| | laboratory tests, SAEs, etc. will be classified by SOC, then sorted |
| | by HLGT, and finally tabulated by PT. |
| | For SOC, the number of patients with a SAE, etc. and the incidence |
| Type of SAE | of SAE, etc. will be listed by SOC internationally agreed order. |
| | For PT, the number and incidence of SAE, etc. will be listed in |
| | ascending order of PT code. |
| | Multiple episodes of the same SAE, etc. (PT) in the same patient |
| | will be tabulated as 1 patient/1 event. |
| | The number of SAE, etc. not related to Zacras will be presented in |
| | parentheses. |

#### (3) Table/figure number

Table 5.9-1

# 5.10 Listing of Occurrence of Serious Adverse Events/Infections in Patients Excluded from Safety Evaluation

(1) Patients included in tabulation/analysis

Patients excluded from safety evaluation

(2) Data tabulated/analyzed

The following variables will be tabulated:

| Variable | Data tabulated/analyzed |
|---------------------------|------------------------------------------------|
| Number of patients with a | Number of patients who experienced a SAE, etc. |
| SAE, etc. | |

| | Ţ |
|---|---|
| | Number of reported SAE, etc. |
| Number of SAE, etc. | Multiple episodes of the same SAE, etc. (PT) in the same patient |
| | will be tabulated as the total number of episodes. |
| | The incidence of SAE, etc. will be calculated as number of patients |
| Incidence of SAE, etc. | with a SAE, etc./number of patients included in safety evaluation × |
| | 100. |
| | SAEs, etc. will be classified by SOC and then tabulated by PT. For |
| | laboratory tests, SAEs, etc. will be classified by SOC, then sorted |
| | by HLGT, and finally tabulated by PT. |
| | For SOC, the number of patients with a SAE, etc. and the incidence |
| | of SAE, etc. will be listed by SOC internationally agreed order. |
| Type of SAE | For PT, the number and incidence of SAE, etc. will be listed in |
| | ascending order of PT code. |
| | Multiple episodes of the same SAE, etc. (PT) in the same patient |
| | will be tabulated as 1 patient/1 event. |
| | The number of SAE, etc. not related to Zacras will be presented in |
| | parentheses. |

Table 5.10-1

#### 5.11 Changes in Test/Measurement Data over Time

#### 5.11.1 Vital Signs (Pulse Rate)

(1) Patients included in tabulation/analysis

Patients included in safety evaluation who have test data at 1 time point or more both before and after treatment with Zacras

(2) Data tabulated/analyzed

For pulse rate (bpm), summary statistics will be calculated for measured values at each time point of measurement [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment]. For the change from the start of treatment with Zacras, summary statistics and 95% CI for the mean will be calculated, and the paired t-test will be performed.

(3) Table/figure number

Table 5.11-1

#### 5.11.2Laboratory Tests

(1) Patients included in tabulation/analysis

Patients included in safety evaluation who have test data at 1 time point or more both before and after treatment with Zacras

(2) Data tabulated/analyzed

For white blood cell count, platelet count, AST, ALT,  $\gamma$ -GTP, serum creatinine, BUN, and serum potassium, summary statistics will be calculated for test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment]. For the change from the start of treatment with Zacras, summary statistics and 95% CI for the mean will be calculated.

(3) Table/figure number

Table 5.11-2

- 5.12 Occurrence of Adverse Drug Reactions/Infections by the Presence or Absence of Concomitant ACE Inhibitor (during the Survey Period)
  - (1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The type of ADR, etc. will be tabulated by the presence or absence of concomitant ACE inhibitor.

The type of ADR, etc. will be tabulated as described in Section 5.1.

A patient with "yes" for concomitant ACE inhibitor (during the survey period) and an ADR, etc. will be handled as a patient with "no" for concomitant ACE inhibitor if the ADR, etc. occurs before the start of concomitant treatment. A patient with "yes" for concomitant

ACE inhibitor (during the survey period) and multiple ADRs, etc. will be handled as a patient with "yes" for concomitant ACE inhibitor if at least one ADR, etc. occurs after the start of concomitant treatment.

(3) Table/figure number

Table 5.12

- 5.13 Occurrence of Adverse Drug Reactions/Infections by the Presence or Absence of Concomitant Aldosterone Antagonist (during the Survey Period)
  - (1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The type of ADR, etc. will be tabulated by the presence or absence of concomitant aldosterone antagonist.

The type of ADR, etc. will be tabulated as described in Section 5.1.

A patient with "yes" for concomitant aldosterone antagonist (during the survey period) and an ADR, etc. will be handled as a patient with "no" for concomitant aldosterone antagonist if the ADR, etc. occurs before the start of concomitant treatment. A patient with "yes" for concomitant aldosterone antagonist (during the survey period) and multiple ADRs, etc. will be handled as a patient with "yes" for concomitant aldosterone antagonist if at least one ADR, etc. occurs after the start of concomitant treatment.

(3) Table/figure number

Table 5.13

- 5.14 Occurrence of Adverse Drug Reactions/Infections by the Presence or Absence of Concomitant Renin Inhibitor (during the Survey Period)
  - (1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The type of ADR, etc. will be tabulated by the presence or absence of concomitant renin inhibitor.

The type of ADR, etc. will be tabulated as described in Section 5.1.

A patient with "yes" for concomitant renin inhibitor (during the survey period) and an ADR, etc. will be handled as a patient with "no" for concomitant renin inhibitor if the ADR, etc. occurs before the start of concomitant treatment. A patient with "yes" for concomitant renin inhibitor (during the survey period) and multiple ADRs, etc. will be handled as a patient with "yes" for concomitant renin inhibitor if at least one ADR, etc. occurs after the start of

concomitant treatment.

(3) Table/figure number

Table 5.14

- 5.15 Occurrence of Adverse Drug Reactions/Infections by the Presence or Absence of Concomitant Diuretic (during the Survey Period)
  - (1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The type of ADR, etc. will be tabulated by the presence or absence of concomitant diuretic.

The type of ADR, etc. will be tabulated as described in Section 5.1.

A patient with "yes" for concomitant diuretic (during the survey period) and an ADR, etc. will be handled as a patient with "no" for concomitant diuretic if the ADR, etc. occurs before the start of concomitant treatment. A patient with "yes" for concomitant diuretic (during the survey period) and multiple ADRs, etc. will be handled as a patient with "yes" for concomitant diuretic if at least one ADR, etc. occurs after the start of concomitant treatment.

(3) Table/figure number

Table 5.15

- 5.16 Occurrence of Adverse Drug Reactions/Infections by the Presence or Absence of Concomitant HCTZ (during the Survey Period)
  - (1) Patients included in tabulation/analysis

Patients included in safety evaluation

(2) Data tabulated/analyzed

The type of ADR, etc. will be tabulated by the presence or absence of concomitant HCTZ.

The type of ADR, etc. will be tabulated as described in Section 5.1.

A patient with "yes" for concomitant HCTZ (during the survey period) and an ADR, etc. will be handled as a patient with "no" for concomitant HCTZ if the ADR, etc. occurs before the start of concomitant treatment. A patient with "yes" for concomitant HCTZ (during the survey period) and multiple ADRs, etc. will be handled as a patient with "yes" for concomitant HCTZ if at least one ADR, etc. occurs after the start of concomitant treatment.

(3) Table/figure number

Table 5.16

#### 6.0 Tabulation/Analysis of Efficacy

#### 6.1 Changes in Blood Pressure over Time

(1) Patients included in tabulation/analysis

Patients included in efficacy evaluation

#### (2) Data tabulated/analyzed

For systolic and diastolic blood pressure, summary statistics will be calculated for test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment]. For the change from the start of treatment with Zacras, summary statistics and 95% CI for the mean will be calculated, and the paired t-test will be performed. In addition, line graph with the mean  $\pm$  standard deviation of test data on the vertical axis and the time point of test on the horizontal axis, and bar graph with the change on the vertical axis and the time point of test on the horizontal axis will be prepared. Paired t-test results will be displayed with an asterisk in graphs.

(3) Table/figure number

Table 6.1, Figure 6.1

#### 6.2 Changes in Blood Pressure over Time <Male>

(1) Patients included in tabulation/analysis

Patients included in efficacy evaluation

(2) Data tabulated/analyzed

For systolic and diastolic blood pressure, test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment] will be tabulated with the stratification factor [sex: male] as described in Section 6.1.

(3) Table/figure number

Table 6.2, Figure 6.2

#### 6.3 Changes in Blood Pressure over Time <Female>

(1) Patients included in tabulation/analysis

Patients included in efficacy evaluation

(2) Data tabulated/analyzed

For systolic and diastolic blood pressure, test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment] will be tabulated with the stratification factor [sex: female] as described in Section 6.1.

(3) Table/figure number

Table 6.3, Figure 6.3

#### 6.4 Changes in Blood Pressure over Time <<65 Years>

(1) Patients included in tabulation/analysis

Patients included in efficacy evaluation

(2) Data tabulated/analyzed

For systolic and diastolic blood pressure, test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment] will be tabulated with the stratification factor [age: <65 years] as described in Section 6.1.

(3) Table/figure number

Table 6.4, Figure 6.4

- 6.5 Changes in Blood Pressure over Time <65 to 74 Years>
  - (1) Patients included in tabulation/analysis

Patients included in efficacy evaluation

(2) Data tabulated/analyzed

For systolic and diastolic blood pressure, test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment] will be tabulated with the stratification factor [age: 65 to 74 years] as described in Section 6.1.

(3) Table/figure number

Table 6.5, Figure 6.5

- 6.6 Changes in Blood Pressure over Time <≥75 Years>
  - (1) Patients included in tabulation/analysis

Patients included in efficacy evaluation

(2) Data tabulated/analyzed

For systolic and diastolic blood pressure, test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment] will be tabulated with the stratification factor [age:  $\geq$ 75 years] as described in Section 6.1.

(3) Table/figure number

Table 6.6, Figure 6.6

- 6.7 Changes in Blood Pressure over Time < Presence or Absence of Concurrent Hepatic Impairment (No)>
  - (1) Patients included in tabulation/analysis

Patients included in efficacy evaluation

(2) Data tabulated/analyzed

For systolic and diastolic blood pressure, test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment] will be tabulated with the stratification factor [presence or absence of concurrent hepatic impairment: no] as described in Section 6.1.

(3) Table/figure number

Table 6.7, Figure 6.7

- 6.8 Changes in Blood Pressure over Time < Presence or Absence of Concurrent Hepatic Impairment (Yes)>
  - (1) Patients included in tabulation/analysis

Patients included in efficacy evaluation

(2) Data tabulated/analyzed

For systolic and diastolic blood pressure, test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment] will be tabulated with the stratification factor [presence or absence of concurrent hepatic impairment: yes] as described in Section 6.1.

(3) Table/figure number

Table 6.8, Figure 6.8

- 6.9 Changes in Blood Pressure over Time < Presence or Absence of Concurrent Renal Impairment (No)>
  - (1) Patients included in tabulation/analysis

Patients included in efficacy evaluation

(2) Data tabulated/analyzed

For systolic and diastolic blood pressure, test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment] will be tabulated with the stratification factor [presence or absence of concurrent renal impairment: no] as described in Section 6.1.

(3) Table/figure number

Table 6.9, Figure 6.9

- 6.10 Changes in Blood Pressure over Time < Presence or Absence of Concurrent Renal Impairment (Yes)>
  - (1) Patients included in tabulation/analysis

Patients included in efficacy evaluation

(2) Data tabulated/analyzed

For systolic and diastolic blood pressure, test data at each time point of test [at the start of

treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment] will be tabulated with the stratification factor [presence or absence of concurrent renal impairment: yes] as described in Section 6.1.

(3) Table/figure number

Table 6.10, Figure 6.10

- 6.11 Changes in Blood Pressure over Time < Concomitant Treatment with Zacras HD/HCTZ 6.25 mg (at the Start of Treatment with Zacras)>
  - (1) Patients included in tabulation/analysis

Patients included in efficacy evaluation

(2) Data tabulated/analyzed

For systolic and diastolic blood pressure, test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment] will be tabulated with the stratification factor [concomitant treatment with Zacras HD/HCTZ 6.25 mg (at the start of treatment with Zacras)] as described in Section 6.1.

(3) Table/figure number

Table 6.11, Figure 6.11

- 6.12 Changes in Blood Pressure over Time <Concomitant Treatment with Zacras HD/HCTZ 12.5 mg (at the Start of Treatment with Zacras)>
  - (1) Patients included in tabulation/analysis

Patients included in efficacy evaluation

(2) Data tabulated/analyzed

For systolic and diastolic blood pressure, test data at each time point of test [at the start of treatment with Zacras, from 1 to 12 months of treatment with Zacras, and at the final assessment] will be tabulated with the stratification factor [concomitant treatment with Zacras HD/HCTZ 12.5 mg (at the start of treatment with Zacras)] as described in Section 6.1.

(3) Table/figure number

Table 6.12, Figure 6.12

- 6.13 Proportion of Patients with Normal Blood Pressure
  - (1) Patients included in tabulation/analysis

Patients included in efficacy evaluation

(2) Data tabulated/analyzed

The proportion of patients with normal blood pressure at the start of the survey and the final assessment will be tabulated.

A patient with normal blood pressure is defined as a patient meeting both of the following criteria:

- •Systolic blood pressure <140 mmHg
- •Diastolic blood pressure <90 mmHg
- (3) Table/figure number

Table 6.13

#### 6.14 Factors that May Affect the Efficacy

(1) Patients included in tabulation/analysis

Patients included in safety evaluation

#### (2) Data tabulated/analyzed

For the changes in systolic and diastolic blood pressure at the final assessment, summary statistics and 95% CI for the mean will be calculated by the variables listed below, and the paired t-test will be performed.

| Variable | Category |
|---|---|
| Sex | Male, female |
| Age | <65 years, ≥65 years |
| | <65 years, 65 to 74 years, ≥75 years |
| Predisposition to hypersensitivity | No, yes, unknown |
| Concurrent illness | No, yes |
| Disposition (multiple tabulation) | Diabetes, dyslipidemia, hyperuricemia, cardiac failure, coronary artery disease (myocardial infarction (including old myocardial infarction), angina, or other), atrial fibrillation, renal impairment (chronic kidney disease (CKD) [diabetic nephropathy, nephrosclerosis, or other] or other), hepatic impairment (hepatic steatosis, alcoholic hepatopathy, or other), cerebrovascular disorder |
| Medical history | No, yes, unknown |
| Body weight (kg) | <40, 40 to <50, 50 to <60, 60 to <70, ≥70, not measured |
| BMI (kg/m <sup>2</sup> ) | <18.5, 18.5 to <25.0, 25.0 to <30.0, ≥30.0, unknown |
| Initial dose of Zacras | LD, HD |
| Presence or absence of change in daily dose of Zacras | No, yes |
| Disposition (multiple tabulation) | $LD \rightarrow HD, HD \rightarrow LD$ |
| Duration of treatment | 1 to 180 days, 181 to 360 days, ≥361 days |
| with Zacras | The denominator is the number of patients treated with Zacras for 1 |

| | day or more to calculate the incidence of AE, etc. for "1 to x days" and the number of patients treated with Zacras for $x + 1$ days or more to calculate the incidence of AE, etc. for " $x + 1$ to y days." |
|---|---|
| Treatment with antihypertensive other than Zacras (at the start of treatment with Zacras) | No, yes |
| Disposition (multiple tabulation)* | ACE inhibitor, ARB, diuretic (thiazide and thiazide analogue diuretic), Ca antagonist, direct renin inhibitor, aldosterone antagonist, potassium-sparing diuretic, fixed-dose combination: ARB + diuretic, fixed-dose combination: ARB + Ca antagonist, fixed-dose combination: calcium antagonist + statin, other |
| Treatment with antihypertensive other than Zacras (during the survey period) | No, yes |
| Disposition (multiple tabulation)* | ACE inhibitor, ARB, diuretic (thiazide and thiazide analogue diuretic), Ca antagonist, direct renin inhibitor, aldosterone antagonist, potassium-sparing diuretic, fixed-dose combination: ARB + diuretic, fixed-dose combination: ARB + Ca antagonist, fixed-dose combination: calcium antagonist + statin, other |
| Treatment with antihypertensive other than Zacras (within 2 months before the start of treatment with Zacras) | No, yes |
| Disposition (multiple tabulation)* | ACE inhibitor, ARB, diuretic (thiazide and thiazide analogue diuretic), Ca antagonist, direct renin inhibitor, aldosterone antagonist, potassium-sparing diuretic, fixed-dose combination: ARB + diuretic, fixed-dose combination: ARB + Ca antagonist, fixed-dose combination: calcium antagonist + statin, other |
| Concomitant non-antihypertensive drug (during the survey period) | No, yes |

| Disposition | |
|---|---|
| (multiple tabulation) | Antidiabetic, antidyslipidemic, antihyperuricemic, other |

\* For fixed-dose combinations, individual ingredients will be tabulated separately. If "fixed-dose combination: ARB + diuretic" is used concomitantly, for instance, "ARB" and "diuretic" will also be tabulated.

# (3) Table/figure number

Table 6.14